CLINICAL TRIAL: NCT02052739
Title: An Open-Label Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of SAGE-547 Injection as Adjunctive Therapy for the Treatment of Super-Refractory Status Epilepticus
Brief Title: Study to Evaluate SAGE-547 Injection as Adjunctive Therapy for the Treatment of Super-Refractory Status Epilepticus
Acronym: SRSE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 547-SSE-201
Record Dates: First submitted 2014-01-28; First posted 2014-02-03 (Estimated); Results first posted 2022-05-03 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2022-04

CONDITIONS: Super-refractory Status Epilepticus
Keywords: Status Epilepticus; Refractory status epilepticus; Super-refractory status epilepticus; SAGE-547; SAGE; Sage Therapeutics
MeSH Terms: conditions — Status Epilepticus | interventions — brexanolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SAGE-547 Standard Dose (Experimental): Participants received SAGE-547 IV loading infusion of 286.6 micrograms per kilogram per hour (μg/kg/hr) for 1 hour on Day 1 followed by maintenance infusion of 86 μg/kg/hr for next 95 hours from Days 1 to 4 (i.e. up to Hour 96) followed by taper infusions of 64.5 μg/kg/hr, 43.0 μg/kg/hr, 21.5 μg/kg/hr at a duration of 8 hours each, on Day 5.
  Interventions: Drug: SAGE-547
- SAGE-547 High Dose (Experimental): Participants received SAGE-547 IV loading infusion of 286.6 μg/kg/hr for 1 hour on Day 1 followed by maintenance infusion A of SAGE-547 86 μg/kg/hr for 23 hours on Day 1 followed by maintenance infusion B of SAGE-547 156 μg/kg/hr for 72 hours from Days 2 to 4 followed by taper infusions of 125 μg/kg/hr, 94 μg/kg/hr, 62 μg/kg/hr, 31 μg/kg/hr at a duration of 6 hours each, on Day 5.
  Interventions: Drug: SAGE-547

INTERVENTIONS:
Drug: SAGE-547 — Solution for injection for IV infusion

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of SAGE-547 in participants in super-refractory status epilepticus (SRSE).

DETAILED DESCRIPTION:
This is an open-label study consisting of a screening period (1 day), 4-day treatment period (96 hours) followed by a 1-day dose taper period (24 hours), a 2-day acute follow-up period, and a 3 week extended follow-up period.

On Day 1 of treatment SRSE participants under seizure suppression or burst-suppression with a continuous intravenous (IV) anti-epileptic drug (AED) (third-line agent) were given a 1-hour IV loading infusion of SAGE-547 followed by a maintenance infusion. After 48 hours of SAGE-547 treatment, the continuous IV AED (third-line agent) was weaned while continuing SAGE-547 at the maintenance infusion for the remainder of the treatment period. After 96 hours (4 days) of therapy with SAGE-547, the dose was to be tapered and discontinued over 24 hours.

The participants would have routine continuous electroencephalogram (EEG) monitoring during the screening period, and continuing until 48 hours after SAGE-547 treatment had completed. Participants would then have follow-up examinations weekly for the next 3 weeks (Days 8, 15, 22, and 29), during which safety and functional assessments would be obtained. Apart from treatment with SAGE-547, all participants would receive the standard of care for adults in SRSE along with ongoing treatment for all underlying medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Participants 2 years of age and older.
* Participants with an EEG-confirmed SRSE diagnosis under concomitant therapy with a continuous IV AED (third-line agent) for ≥ 24 hours. For this study, SRSE is defined by the following criteria and in accordance with those used at major epilepsy treatment centers:

  * Failure to respond to the administration of at least one first-line agent (e.g., benzodiazepine or other emergent initial AED treatment), according to institution standard of care, and
  * Failure to respond to at least one second-line agent (e.g., phenytoin, fosphenytoin, valproate, phenobarbital, levetiracetam or other urgent control AED) according to institution standard of care, and
  * Presence of one or more breakthrough seizures > 6 hours after initiation of the continuous IV AED/third-line agent (e.g., pentobarbital, midazolam, propofol).

Exclusion Criteria:

* Participants with SRSE due to anoxic/hypoxic encephalopathy, children (participants aged less than 18 years) with an encephalopathy due to an underlying progressive neurological disorder.
* Participants with clinically significant electrocardiogram abnormalities.
* Participants with a significant medical or surgical condition that may compromise vital organ systems, or other conditions that would place the participants at increased risk such as dialysis or acute respiratory distress syndrome, severe cardiogenic or vasodilatory shock requiring 2 or more pressors, fulminant hepatic failure, etc.
* Participants who are receiving a continuous IV AED (third-line agent) for seizure suppression or burst-suppression that would require greater than 24 hours to wean.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-03-21 (Actual); Primary Completion 2015-05-03 (Actual); Study Completion 2015-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lasser, MD, MBA, Study Chair — Sage Therapeutics
Locations (16):
- United States (16):
  - Sage Investigational Site, Birmingham, Alabama
  - Sage Investigational Site, Sarasota, Florida
  - Sage Investigational Site, Chicago, Illinois
  - Sage Investigational Site, Wichita, Kansas
  - Sage Investigational Site, New Orleans, Louisiana
  - Sage Investigational Site, Boston, Massachusetts
  - Sage Investigational Site, Ann Arbor, Michigan
  - Sage Investigational Site, Detroit, Michigan
  - Sage Investigational Site, New York, New York
  - Sage Investigational Site, Rochester, New York
  - Sage Investigational Site, Durham, North Carolina
  - Sage Investigational Site, Winston-Salem, North Carolina
  - Sage Investigational Site, Philadelphia, Pennsylvania
  - Sage Investigational Site, Nashville, Tennessee
  - Sage Investigational Site, Dallas, Texas
  - Sage Investigational Site, Temple, Texas

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.

REFERENCES:
- [Background] Rosenthal ES, Claassen J, Wainwright MS, Husain AM, Vaitkevicius H, Raines S, Hoffmann E, Colquhoun H, Doherty JJ, Kanes SJ. Brexanolone as adjunctive therapy in super-refractory status epilepticus. Ann Neurol. 2017 Sep;82(3):342-352. doi: 10.1002/ana.25008. Epub 2017 Sep 11. PMID 28779545
- See also: Sage Therapeutics — http://www.sagerx.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 12 sites in United States from 21 March 2014 to 03 May 2015.
Pre-assignment Details: A total of 25 participants were enrolled into the study to receive either SAGE-547 standard dose or SAGE-547 high dose,19 participants of whom completed the study.
Groups:
- SAGE-547 Standard Dose: Participants received SAGE-547 intravenous (IV) loading infusion of 286.6 micrograms per kilogram per hour (μg/kg/hr) for 1 hour on Day 1 followed by maintenance infusion of 86 μg/kg/hr for next 95 hours from Days 1 to 4 (i.e. up to Hour 96) followed by taper infusions of 64.5 μg/kg/hr, 43.0 μg/kg/hr, 21.5 μg/kg/hr at a duration of 8 hours each, on Day 5.
Period: Overall Study
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Started | 19 | 6
Completed | 14 | 5
Not Completed | 5 | 1
Not completed — Withdrew due to Adverse Event | 3 | 0
Not completed — Participant Died | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who were initiated with an infusion of SAGE-547.
Groups:
- SAGE-547 Standard Dose: Participants received SAGE-547 IV loading infusion of 286.6 μg/kg/hr for 1 hour on Day 1 followed by maintenance infusion of 86 μg/kg/hr for next 95 hours from Days 1 to 4 (i.e. up to Hour 96) followed by taper infusions of 64.5 μg/kg/hr, 43.0 μg/kg/hr, 21.5 μg/kg/hr at a duration of 8 hours each, on Day 5.
- Total: Total of all reporting groups
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose | Total
Number analyzed (Participants) | 19 | 6 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (18.98) | 42.3 (22.11) | 47.6 (19.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 1 | 9
  Male | 11 | 5 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 18 | 5 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 15 | 4 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g., a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. TEAEs are defined as those that begin on or after initiation of the infusion of SAGE-547.
Time Frame: Up to Day 29
Population: Safety population included all participants who were initiated with an infusion of SAGE-547.
Measure: Count of Participants; unit: Participants
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
Participants | 17 | 6

2. Primary Outcome: Change From Baseline (CFB) in National Institutes of Health Stroke Scale (NIH-SS) Total Score
Description: The National Institutes of Health Stroke Scale (NIH-SS) was used to examine the physical and neurological state of the participants. The NIH-SS is a 15-item assessment with measures of level of consciousness, visual gaze and vision loss, facial palsy, motor ability, ataxia, sensory ability, aphasia, dysarthria, and inattention. The total NIHSS score range is from 0 (normal) to 42 (severe impairment), with higher values indicating greater level of neurological impairment.
Time Frame: Baseline (Screening) to infusion at 0-24, 25-48, 49-72, 73-96, 97-120 hours; Acute follow-up at 121-144, 145-168 hours; Extended follow-up at Days 8, 15, 22 and 29
Population: Safety population included all participants who were initiated with an infusion of SAGE-547. Number analyzed is the number of participants with data available for analyses at the given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
score on a scale
  Baseline | 34.2 (4.69) | 33.0 (4.86)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 0-24 hours | 0.7 (2.30) | 0.3 (1.51)
  CFB at Infusion: 25-48 hours | 0.8 (3.47) | -1.5 (6.19)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 49-72 hours | -2.2 (6.70) | -2.3 (4.63)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 73-96 hours | -2.9 (8.08) | -5.5 (6.63)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 17 | 6
  CFB at Infusion: 97-120 hours | -5.6 (7.44) | -6.7 (7.20)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 17 | 6
  CFB at Acute Follow-up: 121-144 hours | -7.0 (8.75) | -10.8 (10.13)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 17 | 4
  CFB at Acute Follow-up: 145-168 hours | -7.5 (9.78) | -12.0 (8.76)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 16 | 5
  CFB at Extended Follow-up: Day 8 | -9.0 (9.54) | -15.4 (11.82)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 16 | 5
  CFB at Extended Follow-up: Day 15 | -16.8 (12.10) | -16.6 (13.30)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 14 | 5
  CFB at Extended Follow-up: Day 22 | -15.1 (14.35) | -17.2 (14.55)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 12 | 5
  CFB at Extended Follow-up: Day 29 | -16.7 (15.34) | -20.6 (13.09)

3. Primary Outcome: Change From Baseline in Vital Sign Parameter: Body Weight
Description: Vital signs included weight, heart rate, blood pressure (systolic blood pressure (SBP) and diastolic blood pressure (DBP)), respiratory rate, temperature, oxygen saturation. CFB in body weight is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
kilograms (kg)
  Baseline | 78.263 (25.3905) | 81.667 (20.3141)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 17 | 6
  CFB at Infusion: 0-24 hours | 0.253 (3.3321) | 0.250 (0.3987)
  CFB at Infusion: 25-48 hours | 1.095 (3.9392) | 1.083 (2.1424)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 49-72 hours | 1.444 (3.5787) | -0.933 (2.9561)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 73-96 hours | 1.517 (4.5509) | -0.033 (4.4275)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 17 | 6
  CFB at Infusion: 97-120 hours | 0.688 (4.3148) | 1.567 (8.8672)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 13 | 6
  CFB at Acute Follow-up: 121-144 hours | -0.631 (6.3734) | 1.650 (12.6751)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 10 | 4
  CFB at Acute Follow-up: 145-168 hours | -0.930 (7.7080) | -5.100 (4.8298)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 11 | 5
  CFB at Extended Follow-up: Day 8 | 0.436 (9.5258) | -1.720 (7.6392)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 12 | 4
  CFB at Extended Follow-up: Day 15 | -0.708 (10.1362) | -6.100 (4.7589)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 9 | 5
  CFB at Extended Follow-up: Day 22 | 0.644 (8.9288) | -3.420 (12.4474)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 8 | 5
  CFB at Extended Follow-up: Day 29 | -6.130 (13.5243) | 0.108 (19.4907)

4. Primary Outcome: Change From Baseline in Vital Sign Parameter: Heart Rate
Description: Vital signs included weight, heart rate, blood pressure (SBP and DBP), respiratory rate, temperature, oxygen saturation. CFB in heart rate is reported in this outcome measure.
Time Frame: Baseline (Screening) to infusion at 0-24 hours: Loading-predose and at 15,30,45 minutes;1,2,4,8 and 24 hour;25-48: 48 hour;49-72:72 hours;73-96: 96 hour;97-120:120 hours;Acute follow-up at 121-144,145-168 hours; Extended Follow-up at Days 8, 15, 22 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: beats per minute (beats/min)
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
beats per minute (beats/min)
  Baseline: number analyzed (Participants) | 18 | 5
  Baseline | 89.3 (14.33) | 81.8 (20.90)
  CFB at Infusion: 0-24 hours: Loading - Pre-Dose: number analyzed (Participants) | 4 | 2
  CFB at Infusion: 0-24 hours: Loading - Pre-Dose | -2.3 (4.65) | -0.5 (2.12)
  CFB at Infusion: 0-24 hours: Loading - 15 minutes: number analyzed (Participants) | 19 | 5
  CFB at Infusion: 0-24 hours: Loading - 15 minutes | -0.7 (3.36) | 0.6 (1.52)
  CFB at Infusion: 0-24 hours: Loading - 30 minutes: number analyzed (Participants) | 19 | 5
  CFB at Infusion: 0-24 hours: Loading - 30 minutes | 0.2 (5.26) | -2.0 (2.45)
  CFB at Infusion: 0-24 hours: Loading - 45 minutes: number analyzed (Participants) | 19 | 5
  CFB at Infusion: 0-24 hours: Loading - 45 minutes | -0.9 (3.98) | -3.6 (4.10)
  CFB at Infusion: 0-24 hours: 1 hour | -1.3 (4.18) | -4.7 (7.26)
  CFB at Infusion: 0-24 hours: 2 hours | -1.6 (4.92) | -0.5 (7.56)
  CFB at Infusion: 0-24 hours: 4 hours | -0.6 (7.65) | -2.8 (8.52)
  CFB at Infusion: 0-24 hours: 8 hours | -3.5 (9.87) | -10.7 (10.07)
  CFB at Infusion: 0-24 hours: 24 hours | -2.2 (13.52) | 1.8 (7.11)
  CFB at Infusion: 25-48 hours: 48 hours | 1.9 (15.09) | -4.8 (8.04)
  CFB at Infusion: 49-72 hours: 72 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 49-72 hours: 72 hours | 5.4 (13.65) | 2.7 (12.42)
  CFB at Infusion: 73-96 hours: 96 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 73-96 hours: 96 hours | 6.8 (14.03) | 8.0 (14.38)
  CFB at Infusion: 97-120 hours: 120 hours: number analyzed (Participants) | 17 | 6
  CFB at Infusion: 97-120 hours: 120 hours | 12.9 (13.43) | 10.7 (28.86)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 17 | 5
  CFB at Acute Follow-up: 121-144 hours | 10.1 (13.10) | 18.0 (23.33)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 17 | 5
  CFB at Acute Follow-up: 145-168 hours | 10.9 (15.77) | 14.8 (17.17)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 16 | 5
  CFB at Extended Follow-up: Day 8 | 11.8 (12.69) | 5.6 (15.34)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 16 | 5
  CFB at Extended Follow-up: Day 15 | 12.8 (15.66) | 6.0 (12.63)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 12 | 5
  CFB at Extended Follow-up: Day 22 | 13.3 (11.92) | 13.6 (27.88)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 10 | 5
  CFB at Extended Follow-up: Day 29 | 9.5 (16.19) | 11.2 (26.54)

5. Primary Outcome: Change From Baseline in Vital Sign Parameter: Blood Pressure - SBP and DBP
Description: Vital signs included weight, heart rate, blood pressure (SBP and DBP), respiratory rate, temperature, oxygen saturation. CFB in SBP and DBP is reported in this outcome measure.
Time Frame: Baseline (Screening) to infusion at 0-24 hours:Loading-predose and at 15,30,45 minutes;1,2,4,8 and 24 hour;25-48: 48 hour;49-72: 72 hour;73-96: 96 hour;97-120:120 hour;Acute follow-up at 121-144,145-168 hours;Extended follow-up at Days 8,15,22 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
millimeters of mercury (mmHg)
  SBP Baseline: number analyzed (Participants) | 18 | 5
  SBP Baseline | 111.1 (14.55) | 111.8 (7.46)
  SBP CFB at Infusion: 0-24 hours: Loading - Pre-Dose: number analyzed (Participants) | 4 | 2
  SBP CFB at Infusion: 0-24 hours: Loading - Pre-Dose | 1.3 (13.23) | 20.0 (28.28)
  SBP CFB at Infusion: 0-24 hours: Loading - 15 minutes: number analyzed (Participants) | 19 | 5
  SBP CFB at Infusion: 0-24 hours: Loading - 15 minutes | -3.2 (8.36) | 5.0 (11.85)
  SBP CFB at Infusion: 0-24 hours: Loading - 30 minutes: number analyzed (Participants) | 19 | 5
  SBP CFB at Infusion: 0-24 hours: Loading - 30 minutes | -4.3 (12.64) | 3.8 (11.12)
  SBP CFB at Infusion: 0-24 hours: Loading - 45 minutes: number analyzed (Participants) | 19 | 5
  SBP CFB at Infusion: 0-24 hours: Loading - 45 minutes | -5.3 (12.55) | -9.4 (12.22)
  SBP CFB at Infusion: 0-24 hours: 1 hour | -7.4 (11.96) | -6.8 (11.39)
  SBP CFB at Infusion: 0-24 hours: 2 hours | -6.1 (15.96) | -5.7 (19.72)
  SBP CFB at Infusion: 0-24 hours: 4 hours | -1.1 (14.40) | -1.7 (11.81)
  SBP CFB at Infusion: 0-24 hours: 8 hours | -5.1 (18.55) | -1.3 (18.02)
  SBP CFB at Infusion: 0-24 hours: 24 hour | -5.6 (19.26) | 5.7 (17.63)
  SBP CFB at Infusion: 25-48 hours: 48 hours | -3.1 (21.49) | 2.5 (21.55)
  SBP CFB at Infusion: 49-72 hours: 72 hours: number analyzed (Participants) | 18 | 6
  SBP CFB at Infusion: 49-72 hours: 72 hours | -2.1 (27.72) | 3.0 (23.83)
  SBP CFB at Infusion: 73-96 hours: 96 hours: number analyzed (Participants) | 18 | 6
  SBP CFB at Infusion: 73-96 hours: 96 hours | 6.2 (24.06) | 11.8 (24.39)
  SBP CFB at Infusion: 97-120 hours: 120 hours: number analyzed (Participants) | 17 | 6
  SBP CFB at Infusion: 97-120 hours: 120 hours | -6.9 (22.13) | -1.8 (21.04)
  SBP CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 17 | 5
  SBP CFB at Acute Follow-up: 121-144 hours | -2.2 (18.67) | 12.8 (21.58)
  SBP CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 17 | 5
  SBP CFB at Acute Follow-up: 145-168 hours | -0.2 (24.46) | 7.0 (25.93)
  SBP CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 16 | 5
  SBP CFB at Extended Follow-up: Day 8 | -0.9 (21.12) | 5.0 (16.02)
  SBP CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 16 | 5
  SBP CFB at Extended Follow-up: Day 15 | 8.9 (19.55) | 3.2 (11.52)
  SBP CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 12 | 5
  SBP CFB at Extended Follow-up: Day 22 | 1.6 (27.60) | 7.0 (6.75)
  SBP CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 10 | 5
  SBP CFB at Extended Follow-up: Day 29 | 2.0 (24.20) | 2.8 (19.77)
  DBP Baseline: number analyzed (Participants) | 18 | 5
  DBP Baseline | 59.7 (8.51) | 60.8 (10.69)
  DBP CFB at Infusion: 0-24 hours: Loading - Pre-Dose: number analyzed (Participants) | 4 | 2
  DBP CFB at Infusion: 0-24 hours: Loading - Pre-Dose | 1.3 (10.53) | 7.5 (10.61)
  DBP CFB at Infusion: 0-24 hours: Loading - 15 minutes: number analyzed (Participants) | 19 | 5
  DBP CFB at Infusion: 0-24 hours: Loading - 15 minutes | -2.1 (5.83) | 2.2 (4.15)
  DBP CFB at Infusion: 0-24 hours: Loading - 30 minutes: number analyzed (Participants) | 19 | 5
  DBP CFB at Infusion: 0-24 hours: Loading - 30 minutes | -2.6 (10.38) | 3.6 (5.41)
  DBP CFB at Infusion: 0-24 hours: Loading - 45 minutes: number analyzed (Participants) | 19 | 5
  DBP CFB at Infusion: 0-24 hours: Loading - 45 minutes | -3.3 (6.26) | -3.6 (7.33)
  DBP CFB at Infusion: 0-24 hours: 1 hour | -3.4 (8.17) | -1.8 (3.25)
  DBP CFB at Infusion: 0-24 hours: 2 hours | -2.8 (6.70) | -3.2 (9.56)
  DBP CFB at Infusion: 0-24 hours: 4 hours | -1.7 (7.36) | 0.0 (8.67)
  DBP CFB at Infusion: 0-24 hours: 8 hours | -2.5 (7.11) | -5.0 (12.17)
  DBP CFB at Infusion: 0-24 hours: 24 hours | -2.9 (12.61) | 6.3 (24.99)
  DBP CFB at Infusion: 25-48 hours: 48 hours | -2.9 (9.01) | -4.0 (7.87)
  DBP CFB at Infusion: 49-72 hours: 72 hours: number analyzed (Participants) | 18 | 6
  DBP CFB at Infusion: 49-72 hours: 72 hours | -1.2 (16.37) | -4.2 (5.42)
  DBP CFB at Infusion: 73-96 hours: 96 hours: number analyzed (Participants) | 18 | 6
  DBP CFB at Infusion: 73-96 hours: 96 hours | 1.1 (12.09) | 3.3 (7.58)
  DBP CFB at Infusion: 97-120 hours: 120 hours: number analyzed (Participants) | 17 | 6
  DBP CFB at Infusion: 97-120 hours: 120 hours | -3.4 (12.65) | 1.0 (12.13)
  DBP CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 17 | 5
  DBP CFB at Acute Follow-up: 121-144 hours | -1.8 (11.53) | 6.6 (8.99)
  DBP CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 17 | 5
  DBP CFB at Acute Follow-up: 145-168 hours | 0.8 (18.15) | 3.0 (18.59)
  DBP CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 16 | 5
  DBP CFB at Extended Follow-up: Day 8 | 1.1 (12.40) | 1.0 (10.89)
  DBP CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 16 | 5
  DBP CFB at Extended Follow-up: Day 15 | 7.9 (11.13) | 4.8 (6.22)
  DBP CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 12 | 5
  DBP CFB at Extended Follow-up: Day 22 | 7.3 (14.67) | 13.4 (11.72)
  DBP CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 10 | 5
  DBP CFB at Extended Follow-up: Day 29 | 7.9 (11.02) | 12.4 (22.78)

6. Primary Outcome: Change From Baseline in Vital Sign Parameter: Respiratory Rate
Description: Vital signs included weight, heart rate, blood pressure (SBP and DBP), respiratory rate, temperature, oxygen saturation. CFB in respiratory rate is reported in this outcome measure.
Time Frame: Baseline (Screening) to infusion at 0-24 hours:Loading-predose and at 15,30,45 minutes;1,2,4,8 and 24 hour;25-48: 48 hour;49-72:72 hours;73-96: 96 hour;97-120:120 hours;Acute follow-up at 121-144,145-168 hours;Extended follow-up at Days 8, 15, 22 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: breaths per min (breaths/min)
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
breaths per min (breaths/min)
  Baseline: number analyzed (Participants) | 18 | 5
  Baseline | 17.4 (4.66) | 13.4 (3.58)
  CFB at Infusion: 0-24 hours: Loading - Pre-Dose: number analyzed (Participants) | 4 | 2
  CFB at Infusion: 0-24 hours: Loading - Pre-Dose | 0.3 (2.75) | -2.0 (1.41)
  CFB at Infusion: 0-24 hours: Loading - 15 minutes: number analyzed (Participants) | 19 | 5
  CFB at Infusion: 0-24 hours: Loading - 15 minutes | 0.2 (2.39) | -0.6 (0.89)
  CFB at Infusion: 0-24 hours: Loading - 30 minutes: number analyzed (Participants) | 19 | 5
  CFB at Infusion: 0-24 hours: Loading - 30 minutes | -0.3 (3.05) | -1.0 (1.41)
  CFB at Infusion: 0-24 hours: Loading - 45 minutes: number analyzed (Participants) | 19 | 5
  CFB at Infusion: 0-24 hours: Loading - 45 minutes | -0.3 (2.64) | 1.0 (2.65)
  CFB at Infusion: 0-24 hours: 1 hour | 0.2 (2.24) | 0.2 (1.47)
  CFB at Infusion: 0-24 hours: 2 hours | 1.1 (2.78) | 0.8 (1.33)
  CFB at Infusion: 0-24 hours: 4 hours | 0.6 (1.98) | -0.2 (1.33)
  CFB at Infusion: 0-24 hours: 8 hours | -0.5 (2.14) | -0.3 (1.86)
  CFB at Infusion: 0-24 hours: 24 hours | 0.3 (4.08) | 0.7 (1.51)
  CFB at Infusion: 25-48 hours: 48 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 25-48 hours: 48 hours | -0.1 (3.21) | -0.8 (3.66)
  CFB at Infusion: 49-72 hours: 72 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 49-72 hours: 72 hours | 1.6 (3.65) | 1.0 (6.96)
  CFB at Infusion: 73-96 hours: 96 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 73-96 hours: 96 hours | 4.7 (6.87) | 1.2 (6.97)
  CFB at Infusion: 97-120 hours: 120 hours: number analyzed (Participants) | 17 | 6
  CFB at Infusion: 97-120 hours: 120 hours | 2.5 (5.62) | 1.0 (4.90)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 17 | 5
  CFB at Acute Follow-up: 121-144 hours | 3.2 (4.25) | 1.4 (5.77)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 17 | 5
  CFB at Acute Follow-up: 145-168 hours | 4.2 (6.08) | 6.0 (6.32)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 16 | 5
  CFB at Extended Follow-up: Day 8 | 4.3 (5.94) | 0.6 (3.05)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 16 | 5
  CFB at Extended Follow-up: Day 15 | 3.7 (5.87) | 5.0 (6.40)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 12 | 5
  CFB at Extended Follow-up: Day 22 | 4.9 (4.32) | 3.0 (6.00)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 10 | 5
  CFB at Extended Follow-up: Day 29 | 3.5 (6.35) | 5.6 (11.28)

7. Primary Outcome: Change From Baseline in Vital Sign Parameter: Body Temperature
Description: Vital signs included weight, heart rate, blood pressure (SBP and DBP), respiratory rate, temperature, oxygen saturation. CFB in body temperature is reported in this outcome measure.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees Fahrenheit (F)
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
degrees Fahrenheit (F)
  Baseline: number analyzed (Participants) | 18 | 5
  Baseline | 99.21 (1.195) | 98.98 (2.312)
  CFB at Infusion: 0-24 hours: Loading - Pre-Dose: number analyzed (Participants) | 4 | 2
  CFB at Infusion: 0-24 hours: Loading - Pre-Dose | -0.80 (0.883) | -0.30 (0.707)
  CFB at Infusion: 0-24 hours: Loading - 15 minutes: number analyzed (Participants) | 17 | 5
  CFB at Infusion: 0-24 hours: Loading - 15 minutes | -0.38 (0.471) | -0.04 (0.329)
  CFB at Infusion: 0-24 hours: Loading - 30 minutes: number analyzed (Participants) | 17 | 5
  CFB at Infusion: 0-24 hours: Loading - 30 minutes | -0.54 (0.628) | -0.14 (0.371)
  CFB at Infusion: 0-24 hours: Loading - 45 minutes: number analyzed (Participants) | 17 | 5
  CFB at Infusion: 0-24 hours: Loading - 45 minutes | -0.58 (0.662) | -0.32 (0.432)
  CFB at Infusion: 0-24 hours: 1 hour | -0.51 (0.614) | -0.55 (0.468)
  CFB at Infusion: 0-24 hours: 2 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 0-24 hours: 2 hours | -0.44 (0.902) | -0.48 (0.407)
  CFB at Infusion: 0-24 hours: 4 hours: number analyzed (Participants) | 16 | 6
  CFB at Infusion: 0-24 hours: 4 hours | -0.17 (1.269) | -0.47 (0.596)
  CFB at Infusion: 0-24 hours: 8 hours: number analyzed (Participants) | 17 | 6
  CFB at Infusion: 0-24 hours: 8 hours | -0.74 (1.361) | -0.52 (0.985)
  CFB at Infusion: 0-24 hours: 24 hours | -0.20 (1.704) | 0.20 (1.474)
  CFB at Infusion: 25-48 hours: 48 hours | -0.51 (1.467) | -0.47 (1.335)
  CFB at Infusion: 49-72 hours: 72 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 49-72 hours: 72 hours | -0.53 (1.522) | -0.47 (1.296)
  CFB at Infusion: 73-96 hour: 96 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 73-96 hour: 96 hours | -0.32 (1.263) | -0.62 (1.283)
  CFB at Infusion: 97-120 hours: 120 hours: number analyzed (Participants) | 17 | 6
  CFB at Infusion: 97-120 hours: 120 hours | -0.14 (1.230) | -0.92 (1.514)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 17 | 5
  CFB at Acute Follow-up: 121-144 hours | 0.06 (1.360) | -0.16 (1.450)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 17 | 5
  CFB at Acute Follow-up: 145-168 hours | -0.29 (1.896) | -0.20 (0.652)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 16 | 5
  CFB at Extended Follow-up: Day 8 | 0.03 (1.010) | -0.46 (0.684)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 16 | 5
  CFB at Extended Follow-up: Day 15 | -0.44 (1.852) | -0.42 (0.740)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 12 | 5
  CFB at Extended Follow-up: Day 22 | -0.62 (1.834) | -0.96 (1.790)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 9 | 5
  CFB at Extended Follow-up: Day 29 | -0.69 (1.515) | -1.20 (2.164)

8. Primary Outcome: Change From Baseline in Vital Sign Parameter: Oxygen Saturation
Description: Vital signs included weight, heart rate, blood pressure (SBP and DBP), respiratory rate, temperature, oxygen saturation. Oxygen saturation is a measure of how much hemoglobin is currently bound to oxygen compared to how much hemoglobin remains unbound. CFB in oxygen saturation is reported in this outcome measure.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
percentage of oxygen saturation
  Baseline: number analyzed (Participants) | 18 | 5
  Baseline | 98.8 (2.26) | 98.6 (1.67)
  CFB at Infusion: 0-24 hours: Loading - Pre-Dose: number analyzed (Participants) | 4 | 2
  CFB at Infusion: 0-24 hours: Loading - Pre-Dose | 0.0 (0.00) | 0.5 (0.71)
  CFB at Infusion: 0-24 hours: Loading - 15 minutes: number analyzed (Participants) | 19 | 5
  CFB at Infusion: 0-24 hours: Loading - 15 minutes | 0.0 (0.33) | 0.2 (0.45)
  CFB at Infusion: 0-24 hours: Loading - 30 minutes: number analyzed (Participants) | 19 | 5
  CFB at Infusion: 0-24 hours: Loading - 30 minutes | -0.3 (1.45) | 0.4 (1.52)
  CFB at Infusion: 0-24 hours: Loading - 45 minutes: number analyzed (Participants) | 19 | 5
  CFB at Infusion: 0-24 hours: Loading - 45 minutes | -0.2 (1.08) | 0.2 (1.92)
  CFB at Infusion: 0-24 hours: 1 hour | -0.5 (2.48) | 0.0 (1.55)
  CFB at Infusion: 0-24 hours: 2 hours | 0.1 (1.10) | -1.3 (4.76)
  CFB at Infusion: 0-24 hours: 4 hours | -0.2 (0.69) | 1.2 (1.33)
  CFB at Infusion: 0-24 hours: 8 hours | -0.1 (1.45) | 1.0 (0.89)
  CFB at Infusion: 0-24 hours: 24 hours | 0.0 (1.15) | -0.7 (1.75)
  CFB at Infusion: 25-48 hours: 48 hours | -0.6 (2.75) | 0.8 (0.98)
  CFB at Infusion: 49-72 hours: 72 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 49-72 hours: 72 hours | -0.1 (2.01) | 0.3 (1.97)
  CFB at Infusion: 73-96 hours: 96 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 73-96 hours: 96 hours | -0.3 (2.95) | -0.8 (2.48)
  CFB at Infusion: 97-120 hours: 120 hours: number analyzed (Participants) | 17 | 6
  CFB at Infusion: 97-120 hours: 120 hours | -0.5 (2.62) | -1.3 (2.34)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 17 | 5
  CFB at Acute Follow-up: 121-144 hours | 0.1 (2.11) | 0.0 (1.58)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 17 | 5
  CFB at Acute Follow-up: 145-168 hours | -0.3 (2.31) | -0.8 (2.86)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 16 | 5
  CFB at Extended Follow-up: Day 8 | -0.5 (2.58) | -0.2 (1.64)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 16 | 5
  CFB at Extended Follow-up: Day 15 | -1.1 (2.90) | 0.4 (0.55)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 12 | 5
  CFB at Extended Follow-up: Day 22 | -6.9 (22.32) | 0.6 (1.52)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 9 | 5
  CFB at Extended Follow-up: Day 29 | -1.3 (3.54) | -1.2 (1.30)

9. Primary Outcome: Change From Baseline in Serum Chemistry Parameter: Alanine Aminotransferase Levels
Description: Serum chemistry measures included alanine aminotransferase, albumin, aspartate aminotransferase, bicarbonate, bilirubin, blood urea nitrogen, calcium, chloride, creatine kinase, creatinine, glucose, lipase, magnesium, potassium, protein, sodium. CFB in alanine aminotransferase levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: international units per liter (IU/L)
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
international units per liter (IU/L)
  Baseline | 48.7 (82.92) | 40.0 (32.47)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 17 | 6
  CFB at Infusion: 0-24 hours | 8.2 (23.96) | 17.0 (42.85)
  CFB at Infusion: 25-48 hours: number analyzed (Participants) | 17 | 6
  CFB at Infusion: 25-48 hours | 11.0 (39.62) | 39.3 (69.34)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 16 | 6
  CFB at Infusion: 49-72 hours | 5.6 (42.77) | 36.5 (48.02)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 16 | 6
  CFB at Infusion: 73-96 hours | 1.9 (50.97) | 84.0 (124.28)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 15 | 6
  CFB at Infusion: 97-120 hours | 4.3 (64.93) | 233.3 (475.33)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 14 | 6
  CFB at Acute Follow-up: 121-144 hours | 4.6 (75.63) | 109.5 (222.80)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 14 | 6
  CFB at Acute Follow-up: 145-168 hours | 5.6 (72.25) | 48.5 (107.03)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 14 | 5
  CFB at Extended Follow-up: Day 8 | 4.9 (69.89) | 0.4 (29.80)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 13 | 5
  CFB at Extended Follow-up: Day 15 | -4.5 (85.06) | 32.2 (47.21)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 13 | 4
  CFB at Extended Follow-up: Day 22 | -3.6 (46.91) | 44.0 (65.01)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 10 | 3
  CFB at Extended Follow-up: Day 29 | 61.2 (309.38) | 374.0 (404.96)

10. Primary Outcome: Change From Baseline in Serum Chemistry Parameter: Albumin Levels
Description: Serum chemistry measures included alanine aminotransferase, albumin, aspartate aminotransferase, bicarbonate, bilirubin, blood urea nitrogen, calcium, chloride, creatine kinase, creatinine, glucose, lipase, magnesium, potassium, protein, sodium. CFB in albumin levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
grams per liter (g/L)
  Baseline | 26.7 (4.87) | 21.3 (3.67)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 0-24 hours | -0.3 (1.75) | -1.3 (3.33)
  CFB at Infusion: 25-48 hours | -0.5 (1.84) | -0.7 (7.17)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 49-72 hours | -0.2 (2.32) | 0.7 (5.28)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 73-96 hours | 0.1 (2.26) | 3.8 (8.54)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 17 | 6
  CFB at Infusion: 97-120 hours | -0.1 (2.45) | 5.0 (6.60)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 16 | 6
  CFB at Acute Follow-up: 121-144 hours | 0.3 (2.82) | 5.3 (8.71)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 16 | 6
  CFB at Acute Follow-up: 145-168 hours | 0.6 (3.61) | 7.5 (8.96)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 16 | 5
  CFB at Extended Follow-up: Day 8 | 1.2 (4.34) | 9.2 (9.44)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 16 | 5
  CFB at Extended Follow-up: Day 15 | 2.8 (6.45) | 10.2 (6.22)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 14 | 4
  CFB at Extended Follow-up: Day 22 | 5.7 (7.46) | 9.5 (1.73)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 11 | 3
  CFB at Extended Follow-up: Day 29 | 4.8 (7.91) | 12.3 (4.04)

11. Primary Outcome: Change From Baseline in Serum Chemistry Parameter: Aspartate Aminotransferase Levels
Description: Serum chemistry measures included alanine aminotransferase, albumin, aspartate aminotransferase, bicarbonate, bilirubin, blood urea nitrogen, calcium, chloride, creatine kinase, creatinine, glucose, lipase, magnesium, potassium, protein, sodium. CFB in aspartate aminotransferase levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
IU/L
  Baseline | 43.8 (50.41) | 44.8 (35.87)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 17 | 6
  CFB at Infusion: 0-24 hours | 0.9 (43.24) | 18.3 (31.42)
  CFB at Infusion: 25-48 hours: number analyzed (Participants) | 17 | 6
  CFB at Infusion: 25-48 hours | 7.5 (43.28) | 32.7 (30.66)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 16 | 6
  CFB at Infusion: 49-72 hours | -0.8 (40.40) | 24.5 (24.99)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 16 | 6
  CFB at Infusion: 73-96 hours | 2.4 (39.23) | 146.7 (328.43)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 15 | 6
  CFB at Infusion: 97-120 hours | 8.7 (39.62) | 854.5 (2056.68)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 14 | 6
  CFB at Acute Follow-up: 121-144 hours | 11.8 (35.16) | 440.3 (1067.48)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 14 | 6
  CFB at Acute Follow-up: 145-168 hours | 12.6 (29.27) | 264.7 (654.96)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 14 | 5
  CFB at Extended Follow-up: Day 8 | 10.8 (34.72) | -5.2 (16.63)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 13 | 5
  CFB at Extended Follow-up: Day 15 | 2.9 (33.33) | 29.0 (48.93)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 13 | 4
  CFB at Extended Follow-up: Day 22 | 15.8 (68.73) | 25.0 (55.47)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 10 | 3
  CFB at Extended Follow-up: Day 29 | 24.9 (121.92) | 1888.0 (3115.96)

12. Primary Outcome: Change From Baseline in Serum Chemistry Parameter: Bicarbonate Levels
Description: Serum chemistry measures included alanine aminotransferase, albumin, aspartate aminotransferase, bicarbonate, bilirubin, blood urea nitrogen, calcium, chloride, creatine kinase, creatinine, glucose, lipase, magnesium, potassium, protein, sodium. CFB in bicarbonate levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
millimoles per liter (mmol/L)
  Baseline | 22.29 (5.247) | 24.52 (4.481)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 0-24 hours | 0.29 (2.077) | -0.85 (2.411)
  CFB at Infusion: 25-48 hours | 0.68 (3.607) | -0.90 (2.205)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 17 | 6
  CFB at Infusion: 49-72 hours | 1.12 (3.252) | -0.98 (3.060)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 73-96 hours | 1.10 (3.258) | -0.20 (3.200)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 17 | 6
  CFB at Infusion: 97-120 hours | 1.42 (4.187) | -0.83 (4.262)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 17 | 6
  CFB at Acute Follow-up: 121-144 hours | 1.68 (4.834) | -1.75 (5.511)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 15 | 6
  CFB at Acute Follow-up: 145-168 hours | 1.85 (5.119) | -2.15 (5.829)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 15 | 5
  CFB at Extended Follow-up: Day 8 | 1.27 (5.397) | -0.06 (4.463)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 15 | 5
  CFB at Extended Follow-up: Day 15 | 0.95 (5.309) | 1.14 (6.527)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 13 | 5
  CFB at Extended Follow-up: Day 22 | 1.45 (6.239) | 1.56 (5.447)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 12 | 4
  CFB at Extended Follow-up: Day 29 | 2.59 (6.432) | 0.25 (6.850)

13. Primary Outcome: Change From Baseline in Serum Chemistry Parameter: Bilirubin Levels
Description: Serum chemistry measures included alanine aminotransferase, albumin, aspartate aminotransferase, bicarbonate, bilirubin, blood urea nitrogen, calcium, chloride, creatine kinase, creatinine, glucose, lipase, magnesium, potassium, protein, sodium. CFB in bilirubin levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micromoles per liter (μmol/L)
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
micromoles per liter (μmol/L)
  Baseline | 15.3900 (37.32086) | 6.8400 (7.41438)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 17 | 6
  CFB at Infusion: 0-24 hours | -2.8165 (7.32863) | 0.8550 (2.35707)
  CFB at Infusion: 25-48 hours: number analyzed (Participants) | 17 | 6
  CFB at Infusion: 25-48 hours | -3.0176 (8.68845) | 0.0000 (5.72275)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 16 | 6
  CFB at Infusion: 49-72 hours | -1.0688 (3.11420) | -1.4250 (6.15758)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 16 | 6
  CFB at Infusion: 73-96 hours | 1.9237 (5.14423) | -0.8550 (5.59356)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 15 | 6
  CFB at Infusion: 97-120 hours | 1.3680 (6.27296) | 0.0000 (7.33508)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 14 | 6
  CFB at Acute Follow-up: 121-144 hours | 1.4657 (6.56677) | 0.5700 (9.34522)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 14 | 6
  CFB at Acute Follow-up: 145-168 hours | 3.9086 (10.20347) | 3.7050 (14.56682)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 14 | 5
  CFB at Extended Follow-up: Day 8 | 7.2064 (18.06184) | -2.0520 (7.49284)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 13 | 5
  CFB at Extended Follow-up: Day 15 | 7.6292 (25.00165) | -2.3940 (7.31512)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 13 | 4
  CFB at Extended Follow-up: Day 22 | 4.4197 (18.18369) | -0.4275 (5.10619)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 10 | 3
  CFB at Extended Follow-up: Day 29 | 26.5050 (69.14760) | 2.2800 (1.97454)

14. Primary Outcome: Change From Baseline in Serum Chemistry Parameter: Blood Urea Nitrogen Levels
Description: Serum chemistry measures included alanine aminotransferase, albumin, aspartate aminotransferase, bicarbonate, bilirubin, blood urea nitrogen, calcium, chloride, creatine kinase, creatinine, glucose, lipase, magnesium, potassium, protein, sodium. CFB in blood urea nitrogen levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
mmol/L
  Baseline | 4.7162 (2.04935) | 4.9980 (1.62817)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 0-24 hours | 0.5752 (0.90926) | -0.1785 (0.58661)
  CFB at Infusion: 25-48 hours | 1.2025 (1.55708) | -0.7140 (1.17322)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 49-72 hours | 1.3090 (1.79547) | -0.8925 (1.16778)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 73-96 hours | 1.6462 (2.02001) | -0.1785 (1.99090)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 17 | 6
  CFB at Infusion: 97-120 hours | 2.0160 (2.22925) | 0.6545 (2.82384)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 17 | 6
  CFB at Acute Follow-up: 121-144 hours | 2.1000 (2.37104) | 2.0825 (2.79663)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 16 | 6
  CFB at Acute Follow-up: 145-168 hours | 2.1197 (2.64106) | 1.9040 (2.79890)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 16 | 5
  CFB at Extended Follow-up: Day 8 | 1.8743 (2.74527) | 1.1424 (2.55448)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 16 | 5
  CFB at Extended Follow-up: Day 15 | 1.5396 (2.64507) | 0.0714 (2.14794)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 14 | 5
  CFB at Extended Follow-up: Day 22 | 2.0145 (5.10015) | -0.0714 (3.73914)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 12 | 4
  CFB at Extended Follow-up: Day 29 | 1.0115 (3.40329) | 1.3388 (0.79160)

15. Primary Outcome: Change From Baseline in Serum Chemistry Parameter: Calcium Levels
Description: Serum chemistry measures included alanine aminotransferase, albumin, aspartate aminotransferase, bicarbonate, bilirubin, blood urea nitrogen, calcium, chloride, creatine kinase, creatinine, glucose, lipase, magnesium, potassium, protein, sodium. CFB in calcium levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
mmol/L
  Baseline | 0.2037 (0.01153) | 0.1950 (0.02074)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 0-24 hours | 0.0015 (0.00733) | 0.0021 (0.00732)
  CFB at Infusion: 25-48 hours | 0.0036 (0.00984) | 0.0017 (0.01765)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 49-72 hours | 0.0056 (0.01521) | 0.0067 (0.02149)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 73-96 hours | 0.0078 (0.01522) | 0.0079 (0.02947)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 17 | 6
  CFB at Infusion: 97-120 hours | 0.0084 (0.01714) | 0.0117 (0.02493)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 17 | 6
  CFB at Acute Follow-up: 121-144 hours | 0.0071 (0.01703) | 0.0125 (0.02766)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 16 | 6
  CFB at Acute Follow-up: 145-168 hours | 0.0100 (0.01180) | 0.0092 (0.02553)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 16 | 5
  CFB at Extended Follow-up: Day 8 | 0.0114 (0.01016) | 0.0170 (0.01866)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 16 | 5
  CFB at Extended Follow-up: Day 15 | 0.0172 (0.01873) | 0.0170 (0.01681)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 14 | 4
  CFB at Extended Follow-up: Day 22 | 0.0202 (0.03017) | 0.0219 (0.00688)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 12 | 3
  CFB at Extended Follow-up: Day 29 | 0.0121 (0.02749) | 0.0300 (0.00750)

16. Primary Outcome: Change From Baseline in Serum Chemistry Parameter: Chloride Levels
Description: Serum chemistry measures included alanine aminotransferase, albumin, aspartate aminotransferase, bicarbonate, bilirubin, blood urea nitrogen, calcium, chloride, creatine kinase, creatinine, glucose, lipase, magnesium, potassium, protein, sodium. CFB in chloride levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
mmol/L
  Baseline | 110.0 (6.21) | 109.7 (3.72)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 0-24 hours | 0.2 (2.82) | -3.5 (3.56)
  CFB at Infusion: 25-48 hours | -0.6 (3.32) | -0.5 (5.17)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 49-72 hours | -1.1 (3.74) | 0.5 (6.60)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 73-96 hours | -1.6 (4.22) | -0.3 (4.63)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 17 | 6
  CFB at Infusion: 97-120 hours | -2.9 (5.07) | -2.7 (2.73)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 17 | 6
  CFB at Acute Follow-up: 121-144 hours | -2.5 (6.96) | -1.8 (4.92)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 16 | 6
  CFB at Acute Follow-up: 145-168 hours | -4.1 (7.36) | -1.2 (3.97)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 16 | 5
  CFB at Extended Follow-up: Day 8 | -4.0 (7.32) | -3.4 (5.55)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 16 | 5
  CFB at Extended Follow-up: Day 15 | -5.9 (9.02) | -4.6 (12.12)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 14 | 5
  CFB at Extended Follow-up: Day 22 | -4.1 (8.63) | -10.8 (5.81)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 12 | 4
  CFB at Extended Follow-up: Day 29 | -7.2 (6.73) | -11.0 (4.69)

17. Primary Outcome: Change From Baseline in Serum Chemistry Parameter: Creatine Kinase Levels
Description: Serum chemistry measures included alanine aminotransferase, albumin, aspartate aminotransferase, bicarbonate, bilirubin, blood urea nitrogen, calcium, chloride, creatine kinase, creatinine, glucose, lipase, magnesium, potassium, protein, sodium. CFB in creatine kinase levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
IU/L
  Baseline: number analyzed (Participants) | 16 | 5
  Baseline | 164.6 (297.58) | 1056.4 (1476.88)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 14 | 4
  CFB at Infusion: 0-24 hours | -5.4 (99.29) | 80.0 (343.91)
  CFB at Infusion: 25-48 hours: number analyzed (Participants) | 15 | 4
  CFB at Infusion: 25-48 hours | -41.5 (204.71) | -77.0 (226.45)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 14 | 5
  CFB at Infusion: 49-72 hours | -52.8 (240.39) | -35.2 (375.74)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 13 | 5
  CFB at Infusion: 73-96 hours | -54.8 (250.36) | 187.8 (428.72)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 12 | 5
  CFB at Infusion: 97-120 hours | -69.4 (267.62) | 1034.6 (2557.56)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 11 | 5
  CFB at Acute Follow-up: 121-144 hours | -94.9 (280.01) | 864.2 (2487.87)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 11 | 5
  CFB at Acute Follow-up: 145-168 hours | -43.8 (269.89) | 1462.6 (3745.02)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 11 | 4
  CFB at Extended Follow-up: Day 8 | -39.5 (286.63) | -67.0 (684.14)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 10 | 4
  CFB at Extended Follow-up: Day 15 | -70.5 (293.08) | -294.5 (520.14)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 9 | 2
  CFB at Extended Follow-up: Day 22 | -108.7 (284.99) | -245.5 (217.08)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 7 | 3
  CFB at Extended Follow-up: Day 29 | 5.9 (51.57) | -356.7 (596.58)

18. Primary Outcome: Change From Baseline in Serum Chemistry Parameter: Creatinine Levels
Description: Serum chemistry measures included alanine aminotransferase, albumin, aspartate aminotransferase, bicarbonate, bilirubin, blood urea nitrogen, calcium, chloride, creatine kinase, creatinine, glucose, lipase, magnesium, potassium, protein, sodium. CFB in creatinine levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
μmol/L
  Baseline | 61.8335 (38.35138) | 66.1527 (26.85624)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 0-24 hours | 3.5851 (21.18016) | -4.2727 (3.96981)
  CFB at Infusion: 25-48 hours | -0.3257 (17.04796) | -2.7993 (9.97654)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 49-72 hours | -5.4513 (17.92081) | -5.1567 (13.15250)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 73-96 hours | -9.0364 (24.69353) | 2.6520 (34.21891)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 17 | 6
  CFB at Infusion: 97-120 hours | -11.1800 (28.19797) | 15.1753 (34.57069)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 17 | 6
  CFB at Acute Follow-up: 121-144 hours | -10.4000 (30.51166) | 32.4133 (73.92834)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 16 | 6
  CFB at Acute Follow-up: 145-168 hours | -6.5748 (39.93224) | 37.8647 (103.07822)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 16 | 5
  CFB at Extended Follow-up: Day 8 | -9.8345 (34.60628) | -1.5912 (12.81648)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 16 | 5
  CFB at Extended Follow-up: Day 15 | -7.1825 (30.96420) | -3.3592 (13.75749)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 14 | 5
  CFB at Extended Follow-up: Day 22 | -4.6726 (33.58740) | -11.6688 (33.48365)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 12 | 4
  CFB at Extended Follow-up: Day 29 | 11.7867 (78.66321) | 0.0000 (23.06320)

19. Primary Outcome: Change From Baseline in Serum Chemistry Parameter: Glucose Levels
Description: Serum chemistry measures included alanine aminotransferase, albumin, aspartate aminotransferase, bicarbonate, bilirubin, blood urea nitrogen, calcium, chloride, creatine kinase, creatinine, glucose, lipase, magnesium, potassium, protein, sodium. CFB in glucose levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
mmol/L
  Baseline | 7.0731 (1.60940) | 7.1238 (2.48860)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 0-24 hours | 0.7247 (1.21847) | 2.5905 (3.70841)
  CFB at Infusion: 25-48 hours | 0.2542 (1.75414) | 0.6661 (1.44582)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 49-72 hours | 1.0886 (2.99912) | 1.4155 (3.15690)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 73-96 hours | 0.0956 (1.98021) | 0.2405 (1.85063)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 17 | 6
  CFB at Infusion: 97-120 hours | 0.4539 (1.53147) | 0.2035 (2.89966)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 17 | 6
  CFB at Acute Follow-up: 121-144 hours | 0.1437 (2.20744) | 0.5644 (1.44173)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 16 | 6
  CFB at Acute Follow-up: 145-168 hours | -0.1457 (1.83254) | -0.2683 (1.26456)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 16 | 5
  CFB at Extended Follow-up: Day 8 | -0.1596 (1.85981) | -1.4766 (2.48794)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 16 | 5
  CFB at Extended Follow-up: Day 15 | -0.4788 (1.91895) | -0.0999 (3.18721)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 14 | 5
  CFB at Extended Follow-up: Day 22 | -0.4084 (2.50478) | -0.1554 (4.07581)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 12 | 4
  CFB at Extended Follow-up: Day 29 | -1.1565 (1.79106) | -1.5959 (2.23900)

20. Primary Outcome: Change From Baseline in Serum Chemistry Parameter: Lipase Levels
Description: Serum chemistry measures included alanine aminotransferase, albumin, aspartate aminotransferase, bicarbonate, bilirubin, blood urea nitrogen, calcium, chloride, creatine kinase, creatinine, glucose, lipase, magnesium, potassium, protein, sodium. CFB in lipase levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
IU/L
  Baseline: number analyzed (Participants) | 15 | 3
  Baseline | 69.7 (108.56) | 48.3 (55.19)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 14 | 3
  CFB at Infusion: 0-24 hours | -13.4 (43.77) | 3.3 (3.21)
  CFB at Infusion: 25-48 hours: number analyzed (Participants) | 15 | 3
  CFB at Infusion: 25-48 hours | -7.5 (34.95) | 9.3 (13.58)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 14 | 3
  CFB at Infusion: 49-72 hours | -14.4 (36.77) | 0.0 (1.73)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 14 | 3
  CFB at Infusion: 73-96 hours | -22.4 (64.01) | 18.0 (25.36)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 13 | 3
  CFB at Infusion: 97-120 hours | -20.5 (63.33) | -6.7 (22.74)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 13 | 3
  CFB at Acute Follow-up: 121-144 hours | -20.3 (91.54) | -10.7 (37.87)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 12 | 3
  CFB at Acute Follow-up: 145-168 hours | -11.7 (99.60) | 9.3 (16.92)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 13 | 3
  CFB at Extended Follow-up: Day 8 | -3.7 (100.78) | 37.0 (28.16)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 12 | 3
  CFB at Extended Follow-up: Day 15 | 24.7 (44.42) | 19.7 (100.17)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 10 | 2
  CFB at Extended Follow-up: Day 22 | 14.1 (38.25) | -15.0 (84.85)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 8 | 3
  CFB at Extended Follow-up: Day 29 | -8.3 (35.42) | 0.0 (31.00)

21. Primary Outcome: Change From Baseline in Serum Chemistry Parameter: Magnesium Levels
Description: Serum chemistry measures included alanine aminotransferase, albumin, aspartate aminotransferase, bicarbonate, bilirubin, blood urea nitrogen, calcium, chloride, creatine kinase, creatinine, glucose, lipase, magnesium, potassium, protein, sodium. CFB in magnesium levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
mmol/L
  Baseline | 0.8969 (0.19546) | 0.8607 (0.14418)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 0-24 hours | -0.0219 (0.11853) | -0.0441 (0.06638)
  CFB at Infusion: 25-48 hours | -0.0194 (0.14406) | -0.0319 (0.11737)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 49-72 hours | -0.0430 (0.11666) | -0.0167 (0.12869)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 17 | 6
  CFB at Infusion: 73-96 hours | -0.0374 (0.17268) | 0.0304 (0.16521)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 16 | 6
  CFB at Infusion: 97-120 hours | -0.0151 (0.22358) | 0.0754 (0.10859)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 16 | 6
  CFB at Acute Follow-up: 121-144 hours | -0.0348 (0.18742) | 0.0534 (0.13315)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 16 | 6
  CFB at Acute Follow-up: 145-168 hours | -0.0151 (0.21498) | 0.0519 (0.15865)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 15 | 5
  CFB at Extended Follow-up: Day 8 | -0.0435 (0.15736) | -0.0811 (0.16860)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 14 | 5
  CFB at Extended Follow-up: Day 15 | -0.0645 (0.15320) | -0.0494 (0.09381)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 12 | 4
  CFB at Extended Follow-up: Day 22 | -0.0564 (0.19263) | -0.1264 (0.15097)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 10 | 3
  CFB at Extended Follow-up: Day 29 | -0.1484 (0.28794) | -0.0608 (0.08902)

22. Primary Outcome: Change From Baseline in Serum Chemistry Parameter: Potassium Levels
Description: Serum chemistry measures included alanine aminotransferase, albumin, aspartate aminotransferase, bicarbonate, bilirubin, blood urea nitrogen, calcium, chloride, creatine kinase, creatinine, glucose, lipase, magnesium, potassium, protein, sodium. CFB in potassium levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
mmol/L
  Baseline | 3.76 (0.439) | 3.87 (0.301)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 0-24 hours | 0.01 (0.515) | -0.03 (0.242)
  CFB at Infusion: 25-48 hours | 0.15 (0.717) | -0.10 (0.329)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 49-72 hours | 0.17 (0.788) | -0.37 (1.117)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 73-96 hours | 0.05 (0.651) | 0.22 (0.601)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 17 | 6
  CFB at Infusion: 97-120 hours | 0.00 (0.446) | 0.35 (0.497)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 17 | 6
  CFB at Acute Follow-up: 121-144 hours | -0.02 (0.542) | 0.37 (0.582)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 16 | 6
  CFB at Acute Follow-up: 145-168 hours | -0.06 (0.578) | 0.75 (0.946)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 16 | 5
  CFB at Extended Follow-up: Day 8 | 0.07 (0.585) | 0.10 (0.255)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 16 | 5
  CFB at Extended Follow-up: Day 15 | 0.04 (0.734) | 0.42 (0.657)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 14 | 5
  CFB at Extended Follow-up: Day 22 | 0.12 (0.654) | 0.32 (0.683)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 12 | 4
  CFB at Extended Follow-up: Day 29 | 0.21 (0.442) | 0.38 (0.741)

23. Primary Outcome: Change From Baseline in Serum Chemistry Parameter: Protein Levels
Description: Serum chemistry measures included alanine aminotransferase, albumin, aspartate aminotransferase, bicarbonate, bilirubin, blood urea nitrogen, calcium, chloride, creatine kinase, creatinine, glucose, lipase, magnesium, potassium, protein, sodium. CFB in protein levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
g/L
  Baseline | 56.5 (9.91) | 52.2 (7.52)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 16 | 6
  CFB at Infusion: 0-24 hours | 0.4 (1.71) | 1.0 (5.51)
  CFB at Infusion: 25-48 hours: number analyzed (Participants) | 17 | 6
  CFB at Infusion: 25-48 hours | 1.1 (2.34) | 1.5 (5.92)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 15 | 6
  CFB at Infusion: 49-72 hours | 1.3 (4.08) | 4.0 (6.69)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 16 | 6
  CFB at Infusion: 73-96 hours | 2.5 (4.10) | 6.5 (5.99)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 15 | 6
  CFB at Infusion: 97-120 hours | 2.8 (2.96) | 8.8 (7.41)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 14 | 6
  CFB at Acute Follow-up: 121-144 hours | 2.5 (5.05) | 6.3 (5.89)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 14 | 6
  CFB at Acute Follow-up: 145-168 hours | 4.1 (4.87) | 7.5 (5.05)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 14 | 5
  CFB at Extended Follow-up: Day 8 | 4.3 (5.06) | 5.6 (5.68)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 11 | 5
  CFB at Extended Follow-up: Day 15 | 5.9 (9.21) | 11.0 (6.44)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 13 | 4
  CFB at Extended Follow-up: Day 22 | 6.7 (10.18) | 16.5 (8.19)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 10 | 3
  CFB at Extended Follow-up: Day 29 | 7.1 (11.56) | 20.0 (7.21)

24. Primary Outcome: Change From Baseline in Serum Chemistry Parameter: Sodium Levels
Description: Serum chemistry measures included alanine aminotransferase, albumin, aspartate aminotransferase, bicarbonate, bilirubin, blood urea nitrogen, calcium, chloride, creatine kinase, creatinine, glucose, lipase, magnesium, potassium, protein, sodium. CFB in sodium levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
mmol/L
  Baseline | 140.6 (4.84) | 141.7 (4.84)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 0-24 hours | 0.1 (2.87) | -3.8 (4.12)
  CFB at Infusion: 25-48 hours | 0.7 (4.31) | 0.3 (5.72)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 49-72 hours | 0.4 (3.88) | 1.7 (6.19)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 73-96 hours | 0.4 (3.50) | 1.5 (3.94)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 17 | 6
  CFB at Infusion: 97-120 hours | 0.0 (4.80) | -0.5 (4.04)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 17 | 6
  CFB at Acute Follow-up: 121-144 hours | -0.3 (5.12) | -1.0 (4.60)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 16 | 6
  CFB at Acute Follow-up: 145-168 hours | -1.2 (5.64) | 0.2 (5.85)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 16 | 5
  CFB at Extended Follow-up: Day 8 | -1.8 (5.65) | 0.0 (5.79)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 16 | 5
  CFB at Extended Follow-up: Day 15 | -2.8 (5.51) | -0.4 (7.64)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 14 | 5
  CFB at Extended Follow-up: Day 22 | 0.0 (5.53) | -3.2 (4.32)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 12 | 4
  CFB at Extended Follow-up: Day 29 | -1.8 (6.34) | -4.5 (1.29)

25. Primary Outcome: Change From Baseline in Hematology Parameter: Basophil Levels
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, erythrocytes mean corpuscular hemoglobin concentration, erythrocytes mean corpuscular hemoglobin, erythrocytes mean corpuscular volume, erythrocytes, hematocrit, hemoglobin, leukocytes, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets. CFB in basophil levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^3 cells per microliter(10^3 cells/uL)
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
10^3 cells per microliter(10^3 cells/uL)
  Baseline: number analyzed (Participants) | 11 | 3
  Baseline | 0.031 (0.0509) | 0.037 (0.0321)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 9 | 3
  CFB at Infusion: 0-24 hours | 0.013 (0.0308) | 0.003 (0.0058)
  CFB at Infusion: 25-48 hours: number analyzed (Participants) | 10 | 3
  CFB at Infusion: 25-48 hours | -0.008 (0.0319) | -0.023 (0.0321)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 8 | 3
  CFB at Infusion: 49-72 hours | 0.009 (0.0230) | -0.007 (0.0208)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 9 | 3
  CFB at Infusion: 73-96 hours | 0.013 (0.0433) | -0.013 (0.0115)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 9 | 2
  CFB at Infusion: 97-120 hours | 0.004 (0.0662) | -0.010 (0.0141)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 8 | 3
  CFB at Acute Follow-up: 121-144 hours | 0.033 (0.0369) | 0.087 (0.1848)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 9 | 3
  CFB at Acute Follow-up: 145-168 hours | 0.006 (0.0669) | -0.017 (0.0153)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 9 | 3
  CFB at Extended Follow-up: Day 8 | 0.014 (0.0745) | -0.017 (0.0153)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 9 | 2
  CFB at Extended Follow-up: Day 15 | 0.031 (0.0366) | 0.040 (0.0849)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 7 | 1
  CFB at Extended Follow-up: Day 22 | 0.020 (0.0216) | 0.000
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 6 | 2
  CFB at Extended Follow-up: Day 29 | 0.017 (0.0288) | -0.005 (0.0071)

26. Primary Outcome: Change From Baseline in Hematology Parameter: Basophils to Leukocytes Ratio Reported in Percentage of Cells
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, erythrocytes mean corpuscular hemoglobin concentration, erythrocytes mean corpuscular hemoglobin, erythrocytes mean corpuscular volume, erythrocytes, hematocrit, hemoglobin, leukocytes, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets. CFB in basophils to leukocytes ratio is reported in terms of percentage of cells in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
percentage of cells
  Baseline: number analyzed (Participants) | 2 | 2
  Baseline | 0.50 (0.707) | 0.00 (0.000)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 1 | 1
  CFB at Infusion: 0-24 hours | 0.00 | 0.00
  CFB at Infusion: 25-48 hours: number analyzed (Participants) | 2 | 1
  CFB at Infusion: 25-48 hours | 0.00 (0.000) | 1.00
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 2 | 1
  CFB at Infusion: 49-72 hours | 0.00 (0.000) | 0.00
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 2 | 1
  CFB at Infusion: 73-96 hours | 0.50 (0.707) | 1.00
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 2 | 1
  CFB at Infusion: 97-120 hours | 0.00 (0.000) | 1.00
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 2 | 1
  CFB at Acute Follow-up: 121-144 hours | 0.00 (0.000) | 0.00
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 2 | 1
  CFB at Acute Follow-up: 145-168 hours | 0.00 (0.000) | 0.00
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 2 | 0
  CFB at Extended Follow-up: Day 8 | 0.00 (0.000) |
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 2 | 0
  CFB at Extended Follow-up: Day 15 | -0.50 (0.707) |
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 2 | 1
  CFB at Extended Follow-up: Day 22 | 0.50 (0.707) | 0.00
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 2 | 0
  CFB at Extended Follow-up: Day 29 | 0.00 (0.000) |

27. Primary Outcome: Change From Baseline in Hematology Parameter: Eosinophil Levels
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, erythrocytes mean corpuscular hemoglobin concentration, erythrocytes mean corpuscular hemoglobin, erythrocytes mean corpuscular volume, erythrocytes, hematocrit, hemoglobin, leukocytes, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets. CFB in eosinophils levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
10^3 cells/uL
  Baseline: number analyzed (Participants) | 11 | 3
  Baseline | 0.3364 (0.42711) | 0.7433 (0.20108)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 10 | 3
  CFB at Infusion: 0-24 hours | 0.0580 (0.17813) | -0.2700 (0.24269)
  CFB at Infusion: 25-48 hours: number analyzed (Participants) | 10 | 3
  CFB at Infusion: 25-48 hours | 0.0660 (0.23538) | -0.2333 (0.45654)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 9 | 3
  CFB at Infusion: 49-72 hours | -0.0911 (0.35069) | -0.6467 (0.14189)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 9 | 3
  CFB at Infusion: 73-96 hours | -0.0811 (0.36381) | -0.5867 (0.07095)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 9 | 3
  CFB at Infusion: 97-120 hours | -0.1878 (0.45535) | -0.4200 (0.41940)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 9 | 3
  CFB at Acute Follow-up: 121-144 hours | -0.2211 (0.44552) | -0.5567 (0.16258)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 9 | 3
  CFB at Acute Follow-up: 145-168 hours | -0.1643 (0.42177) | -0.5567 (0.17898)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 9 | 3
  CFB at Extended Follow-up: Day 8 | -0.1056 (0.40423) | -0.5400 (0.17776)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 9 | 2
  CFB at Extended Follow-up: Day 15 | -0.0078 (0.33774) | 0.0100 (0.26870)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 7 | 1
  CFB at Extended Follow-up: Day 22 | -0.0543 (0.42496) | -0.3000
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 7 | 2
  CFB at Extended Follow-up: Day 29 | -0.0229 (0.39982) | -0.5650 (0.33234)

28. Primary Outcome: Change From Baseline in Hematology Parameter: Eosinophils to Leukocytes Ratio Reported in Percentage of Cells
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, erythrocytes mean corpuscular hemoglobin concentration, erythrocytes mean corpuscular hemoglobin, erythrocytes mean corpuscular volume, erythrocytes, hematocrit, hemoglobin, leukocytes, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets. CFB in eosinophils to leukocytes ratio is reported in terms of percentage of cells in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
percentage of cells
  Baseline: number analyzed (Participants) | 2 | 2
  Baseline | 3.00 (0.000) | 3.00 (0.000)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 1 | 1
  CFB at Infusion: 0-24 hours | 5.00 | -2.00
  CFB at Infusion: 25-48 hours: number analyzed (Participants) | 2 | 1
  CFB at Infusion: 25-48 hours | 0.50 (0.707) | 0.00
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 2 | 1
  CFB at Infusion: 49-72 hours | -0.50 (2.121) | 0.00
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 2 | 1
  CFB at Infusion: 73-96 hours | 0.50 (0.707) | -2.00
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 2 | 1
  CFB at Infusion: 97-120 hours | -1.00 (0.000) | -2.00
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 2 | 1
  CFB at Acute Follow-up: 121-144 hours | -1.50 (0.707) | -3.00
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 2 | 1
  CFB at Acute Follow-up: 145-168 hours | -2.00 (1.414) | -3.00
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 2 | 0
  CFB at Extended Follow-up: Day 8 | 0.50 (2.121) |
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 2 | 0
  CFB at Extended Follow-up: Day 15 | 2.00 (1.414) |
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 2 | 1
  CFB at Extended Follow-up: Day 22 | 1.00 (2.828) | -1.00
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 2 | 0
  CFB at Extended Follow-up: Day 29 | 1.50 (0.707) |

29. Primary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin Concentration Levels
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, erythrocytes mean corpuscular hemoglobin concentration, erythrocytes mean corpuscular hemoglobin, erythrocytes mean corpuscular volume, erythrocytes, hematocrit, hemoglobin, leukocytes, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets. CFB in erythrocytes mean corpuscular hemoglobin concentration levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
g/L
  Baseline: number analyzed (Participants) | 19 | 5
  Baseline | 328.4 (12.54) | 322.6 (12.54)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 18 | 5
  CFB at Infusion: 0-24 hours | -1.2 (12.52) | 1.0 (5.66)
  CFB at Infusion: 25-48 hours: number analyzed (Participants) | 19 | 5
  CFB at Infusion: 25-48 hours | -4.7 (10.43) | 10.4 (12.18)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 18 | 5
  CFB at Infusion: 49-72 hours | -3.4 (7.88) | 5.4 (6.19)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 18 | 5
  CFB at Infusion: 73-96 hours | -3.6 (10.00) | 3.6 (6.35)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 17 | 5
  CFB at Infusion: 97-120 hours | -4.1 (9.33) | 1.8 (3.03)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 17 | 5
  CFB at Acute Follow-up: 121-144 hours | -6.1 (10.65) | -0.4 (2.61)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 15 | 5
  CFB at Acute Follow-up: 145-168 hours | -7.6 (10.44) | 0.4 (5.50)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 15 | 4
  CFB at Extended Follow-up: Day 8 | -7.7 (11.07) | -2.3 (9.54)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 15 | 4
  CFB at Extended Follow-up: Day 15 | -5.5 (14.28) | -0.5 (13.77)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 13 | 4
  CFB at Extended Follow-up: Day 22 | -6.9 (18.40) | 11.5 (32.25)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 11 | 4
  CFB at Extended Follow-up: Day 29 | -4.6 (16.10) | -9.3 (7.50)

30. Primary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin Levels
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, erythrocytes mean corpuscular hemoglobin concentration, erythrocytes mean corpuscular hemoglobin, erythrocytes mean corpuscular volume, erythrocytes, hematocrit, hemoglobin, leukocytes, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets. CFB in erythrocytes mean corpuscular hemoglobin levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: femtomoles (fmol)
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
femtomoles (fmol)
  Baseline: number analyzed (Participants) | 19 | 5
  Baseline | 1.8611 (0.17564) | 1.8335 (0.09869)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 18 | 5
  CFB at Infusion: 0-24 hours | 0.0110 (0.04180) | -0.0149 (0.02996)
  CFB at Infusion: 25-48 hours: number analyzed (Participants) | 19 | 5
  CFB at Infusion: 25-48 hours | -0.0134 (0.03603) | 0.0261 (0.09580)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 18 | 5
  CFB at Infusion: 49-72 hours | -0.0097 (0.03719) | 0.0074 (0.03911)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 18 | 5
  CFB at Infusion: 73-96 hours | -0.0107 (0.04378) | -0.0099 (0.02177)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 17 | 5
  CFB at Infusion: 97-120 hours | -0.0164 (0.04034) | 0.0112 (0.03147)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 17 | 5
  CFB at Acute Follow-up: 121-144 hours | -0.0194 (0.03684) | 0.0099 (0.03582)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 15 | 5
  CFB at Acute Follow-up: 145-168 hours | -0.0112 (0.04763) | 0.0161 (0.03662)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 15 | 4
  CFB at Extended Follow-up: Day 8 | -0.0058 (0.04491) | 0.0155 (0.04927)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 15 | 4
  CFB at Extended Follow-up: Day 15 | -0.0087 (0.09182) | 0.0310 (0.07868)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 13 | 4
  CFB at Extended Follow-up: Day 22 | -0.0306 (0.14055) | 0.0729 (0.14436)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 11 | 4
  CFB at Extended Follow-up: Day 29 | -0.0412 (0.11506) | 0.0341 (0.07457)

31. Primary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume Levels
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, erythrocytes mean corpuscular hemoglobin concentration, erythrocytes mean corpuscular hemoglobin, erythrocytes mean corpuscular volume, erythrocytes, hematocrit, hemoglobin, leukocytes, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets. CFB in erythrocytes mean corpuscular volume levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: femtoliters (fL)
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
femtoliters (fL)
  Baseline: number analyzed (Participants) | 19 | 5
  Baseline | 91.36 (7.651) | 91.50 (4.785)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 18 | 5
  CFB at Infusion: 0-24 hours | 0.68 (1.773) | -0.42 (0.950)
  CFB at Infusion: 25-48 hours: number analyzed (Participants) | 19 | 5
  CFB at Infusion: 25-48 hours | 0.65 (2.202) | -0.82 (1.487)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 18 | 6
  CFB at Infusion: 49-72 hours | 0.46 (2.168) | -1.12 (1.314)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 18 | 5
  CFB at Infusion: 73-96 hours | 0.38 (2.202) | -1.04 (1.146)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 17 | 5
  CFB at Infusion: 97-120 hours | 0.47 (2.560) | 0.10 (1.954)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 17 | 5
  CFB at Acute Follow-up: 121-144 hours | 0.70 (2.362) | 0.76 (1.977)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 15 | 5
  CFB at Acute Follow-up: 145-168 hours | 1.60 (3.270) | 0.36 (1.230)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 15 | 4
  CFB at Extended Follow-up: Day 8 | 1.30 (3.507) | 1.08 (1.090)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 15 | 4
  CFB at Extended Follow-up: Day 15 | 1.20 (4.337) | 2.25 (4.124)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 13 | 4
  CFB at Extended Follow-up: Day 22 | 0.29 (5.675) | 0.75 (3.747)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 11 | 4
  CFB at Extended Follow-up: Day 29 | -0.96 (5.315) | 4.27 (1.775)

32. Primary Outcome: Change From Baseline in Hematology Parameter: Erythrocyte Levels
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, erythrocytes mean corpuscular hemoglobin concentration, erythrocytes mean corpuscular hemoglobin, erythrocytes mean corpuscular volume, erythrocytes, hematocrit, hemoglobin, leukocytes, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets. CFB in erythrocyte levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^6 cells per microliter
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
10^6 cells per microliter
  Baseline: number analyzed (Participants) | 19 | 5
  Baseline | 3.261 (0.7152) | 3.406 (0.5297)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 18 | 5
  CFB at Infusion: 0-24 hours | -0.078 (0.3236) | -0.022 (0.1816)
  CFB at Infusion: 25-48 hours: number analyzed (Participants) | 19 | 5
  CFB at Infusion: 25-48 hours | -0.106 (0.4059) | -0.184 (0.2799)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 18 | 5
  CFB at Infusion: 49-72 hours | -0.162 (0.4112) | -0.218 (0.2072)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 18 | 5
  CFB at Infusion: 73-96 hours | -0.175 (0.4261) | -0.132 (0.3041)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 17 | 5
  CFB at Infusion: 97-120 hours | -0.152 (0.3718) | -0.158 (0.5079)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 17 | 5
  CFB at Acute Follow-up: 121-144 hours | -0.259 (0.4001) | -0.256 (0.5786)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 15 | 5
  CFB at Acute Follow-up: 145-168 hours | -0.199 (0.3819) | -0.200 (0.7139)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 15 | 4
  CFB at Extended Follow-up: Day 8 | -0.196 (0.4508) | -0.463 (0.4367)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 15 | 4
  CFB at Extended Follow-up: Day 15 | 0.115 (0.7317) | -0.133 (0.5821)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 13 | 4
  CFB at Extended Follow-up: Day 22 | 0.285 (0.9424) | 0.105 (0.3493)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 11 | 4
  CFB at Extended Follow-up: Day 29 | 0.607 (0.4754) | 0.248 (0.2924)

33. Primary Outcome: Change From Baseline in Hematology Parameter: Hematocrit Levels
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, erythrocytes mean corpuscular hemoglobin concentration, erythrocytes mean corpuscular hemoglobin, erythrocytes mean corpuscular volume, erythrocytes, hematocrit, hemoglobin, leukocytes, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets. CFB in hematocrit levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: proportion of 1.0 (in liters)
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
proportion of 1.0 (in liters)
  Baseline: number analyzed (Participants) | 19 | 5
  Baseline | 0.2955 (0.05601) | 0.3110 (0.05443)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 18 | 5
  CFB at Infusion: 0-24 hours | -0.0042 (0.02561) | -0.0028 (0.01591)
  CFB at Infusion: 25-48 hours: number analyzed (Participants) | 19 | 5
  CFB at Infusion: 25-48 hours | -0.0058 (0.03430) | -0.0192 (0.02013)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 18 | 5
  CFB at Infusion: 49-72 hours | -0.0123 (0.03371) | -0.0238 (0.01487)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 18 | 5
  CFB at Infusion: 73-96 hours | -0.0131 (0.03564) | -0.0142 (0.02860)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 17 | 5
  CFB at Infusion: 97-120 hours | -0.0108 (0.03167) | -0.0160 (0.04813)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 17 | 5
  CFB at Acute Follow-up: 121-144 hours | -0.0209 (0.03369) | -0.0238 (0.05369)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 15 | 5
  CFB at Acute Follow-up: 145-168 hours | -0.0135 (0.03487) | -0.0182 (0.06883)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 15 | 4
  CFB at Extended Follow-up: Day 8 | -0.0142 (0.03823) | -0.0375 (0.04888)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 15 | 4
  CFB at Extended Follow-up: Day 15 | 0.0143 (0.05903) | -0.0058 (0.05967)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 13 | 4
  CFB at Extended Follow-up: Day 22 | 0.0188 (0.06186) | 0.0128 (0.03157)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 11 | 4
  CFB at Extended Follow-up: Day 29 | 0.0516 (0.04241) | 0.0370 (0.02670)

34. Primary Outcome: Change From Baseline in Hematology Parameter: Hemoglobin Levels
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, erythrocytes mean corpuscular hemoglobin concentration, erythrocytes mean corpuscular hemoglobin, erythrocytes mean corpuscular volume, erythrocytes, hematocrit, hemoglobin, leukocytes, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets. CFB in hemoglobin levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
g/L
  Baseline: number analyzed (Participants) | 19 | 5
  Baseline | 97.3 (19.93) | 100.4 (18.28)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 18 | 5
  CFB at Infusion: 0-24 hours | -2.1 (9.96) | -0.8 (5.26)
  CFB at Infusion: 25-48 hours: number analyzed (Participants) | 19 | 5
  CFB at Infusion: 25-48 hours | -3.8 (11.81) | -3.4 (4.77)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 18 | 5
  CFB at Infusion: 49-72 hours | -5.2 (12.37) | -5.8 (4.21)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 18 | 5
  CFB at Infusion: 73-96 hours | -5.8 (12.89) | -4.0 (7.97)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 17 | 5
  CFB at Infusion: 97-120 hours | -5.4 (11.54) | -4.4 (14.99)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 17 | 5
  CFB at Acute Follow-up: 121-144 hours | -8.8 (12.69) | -7.2 (16.75)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 15 | 5
  CFB at Acute Follow-up: 145-168 hours | -6.8 (12.78) | -5.6 (20.67)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 15 | 4
  CFB at Extended Follow-up: Day 8 | -6.7 (14.41) | -12.3 (12.97)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 15 | 4
  CFB at Extended Follow-up: Day 15 | 2.7 (22.10) | -2.0 (18.65)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 13 | 4
  CFB at Extended Follow-up: Day 22 | 3.8 (21.36) | 8.3 (12.58)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 11 | 4
  CFB at Extended Follow-up: Day 29 | 15.3 (14.50) | 9.5 (9.26)

35. Primary Outcome: Change From Baseline in Hematology Parameter: Leukocyte Levels
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, erythrocytes mean corpuscular hemoglobin concentration, erythrocytes mean corpuscular hemoglobin, erythrocytes mean corpuscular volume, erythrocytes, hematocrit, hemoglobin, leukocytes, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets. CFB in leukocyte levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
10^3 cells/uL
  Baseline: number analyzed (Participants) | 19 | 5
  Baseline | 11.383 (4.3503) | 16.538 (8.5348)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 17 | 5
  CFB at Infusion: 0-24 hours | 1.438 (2.5891) | -0.902 (2.4833)
  CFB at Infusion: 25-48 hours: number analyzed (Participants) | 19 | 5
  CFB at Infusion: 25-48 hours | 0.186 (4.5526) | -3.306 (4.7047)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 18 | 5
  CFB at Infusion: 49-72 hours | -0.227 (6.1765) | -3.090 (5.5029)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 18 | 5
  CFB at Infusion: 73-96 hours | -0.577 (7.1508) | -3.798 (5.5846)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 17 | 5
  CFB at Infusion: 97-120 hours | 0.591 (10.3636) | -3.964 (5.3646)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 17 | 5
  CFB at Acute Follow-up: 121-144 hours | -1.002 (8.9938) | -1.306 (7.5940)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 15 | 5
  CFB at Acute Follow-up: 145-168 hours | -0.123 (10.4153) | -1.652 (7.3674)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 15 | 4
  CFB at Extended Follow-up: Day 8 | -1.145 (7.3294) | -2.188 (6.7041)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 15 | 4
  CFB at Extended Follow-up: Day 15 | -1.692 (5.0282) | -6.118 (7.0178)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 13 | 4
  CFB at Extended Follow-up: Day 22 | -1.132 (4.3853) | -7.248 (7.3886)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 11 | 4
  CFB at Extended Follow-up: Day 29 | -0.790 (6.1582) | -5.840 (4.6825)

36. Primary Outcome: Change From Baseline in Hematology Parameter: Lymphocyte Levels
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, erythrocytes mean corpuscular hemoglobin concentration, erythrocytes mean corpuscular hemoglobin, erythrocytes mean corpuscular volume, erythrocytes, hematocrit, hemoglobin, leukocytes, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets. CFB in lymphocyte levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
10^3 cells/uL
  Baseline: number analyzed (Participants) | 11 | 3
  Baseline | 1.791 (0.8043) | 2.323 (0.5193)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 10 | 3
  CFB at Infusion: 0-24 hours | 0.213 (0.8923) | -0.470 (0.2427)
  CFB at Infusion: 25-48 hours: number analyzed (Participants) | 10 | 3
  CFB at Infusion: 25-48 hours | 0.189 (1.3559) | -1.147 (0.9771)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 9 | 3
  CFB at Infusion: 49-72 hours | 0.302 (1.0584) | -0.640 (1.1037)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 9 | 3
  CFB at Infusion: 73-96 hours | 0.200 (1.1580) | -0.780 (0.4358)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 9 | 3
  CFB at Infusion: 97-120 hours | 0.428 (1.1946) | -0.777 (0.6516)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 9 | 3
  CFB at Acute Follow-up: 121-144 hours | 0.152 (0.9193) | -0.987 (1.0040)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 9 | 3
  CFB at Acute Follow-up: 145-168 hours | 0.360 (0.8965) | -1.013 (0.8799)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 9 | 3
  CFB at Extended Follow-up: Day 8 | 0.482 (0.8724) | -0.700 (0.6720)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 9 | 2
  CFB at Extended Follow-up: Day 15 | 0.392 (0.8363) | -1.140 (0.9334)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 7 | 1
  CFB at Extended Follow-up: Day 22 | 0.343 (0.6667) | -2.200
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 7 | 2
  CFB at Extended Follow-up: Day 29 | 0.427 (0.8182) | -0.845 (1.0677)

37. Primary Outcome: Change From Baseline in Hematology Parameter: Lymphocytes to Leukocytes Ratio Reported in Percentage of Cells
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, erythrocytes mean corpuscular hemoglobin concentration, erythrocytes mean corpuscular hemoglobin, erythrocytes mean corpuscular volume, erythrocytes, hematocrit, hemoglobin, leukocytes, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets. CFB in lymphocytes to leukocytes ratio is reported in terms of percentage of cells in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
percentage of cells
  Baseline: number analyzed (Participants) | 3 | 2
  Baseline | 10.67 (7.024) | 6.50 (7.778)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 2 | 1
  CFB at Infusion: 0-24 hours | -1.00 (0.000) | 4.00
  CFB at Infusion: 25-48 hours: number analyzed (Participants) | 2 | 1
  CFB at Infusion: 25-48 hours | -2.50 (2.121) | 8.00
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 3 | 1
  CFB at Infusion: 49-72 hours | 0.67 (5.033) | 10.00
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 2 | 1
  CFB at Infusion: 73-96 hours | -5.50 (4.950) | 6.00
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 2 | 1
  CFB at Infusion: 97-120 hours | -4.50 (6.364) | 8.00
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 2 | 1
  CFB at Acute Follow-up: 121-144 hours | -6.00 (4.243) | 1.00
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 2 | 1
  CFB at Acute Follow-up: 145-168 hours | -6.00 (2.828) | 1.00
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 2 | 0
  CFB at Extended Follow-up: Day 8 | -6.00 (1.414) |
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 2 | 0
  CFB at Extended Follow-up: Day 15 | -3.50 (3.536) |
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 2 | 1
  CFB at Extended Follow-up: Day 22 | 7.00 (4.243) | 11.00
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 2 | 0
  CFB at Extended Follow-up: Day 29 | 0.50 (2.121) |

38. Primary Outcome: Change From Baseline in Hematology Parameter: Monocyte Levels
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, erythrocytes mean corpuscular hemoglobin concentration, erythrocytes mean corpuscular hemoglobin, erythrocytes mean corpuscular volume, erythrocytes, hematocrit, hemoglobin, leukocytes, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets. CFB in monocyte levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
10^3 cells/uL
  Baseline: number analyzed (Participants) | 11 | 3
  Baseline | 0.6182 (0.26966) | 1.2567 (0.83584)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 10 | 3
  CFB at Infusion: 0-24 hours | 0.2720 (0.39137) | 0.3470 (0.83703)
  CFB at Infusion: 25-48 hours: number analyzed (Participants) | 10 | 3
  CFB at Infusion: 25-48 hours | 0.2830 (0.54878) | -0.1200 (1.05399)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 9 | 3
  CFB at Infusion: 49-72 hours | 0.1267 (0.52906) | -0.0667 (0.06110)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 9 | 3
  CFB at Infusion: 73-96 hours | 0.2978 (0.44409) | 0.4533 (0.39068)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 9 | 3
  CFB at Infusion: 97-120 hours | 0.2322 (0.42364) | 0.1300 (0.96016)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 9 | 3
  CFB at Acute Follow-up: 121-144 hours | 0.2856 (0.47710) | -0.1400 (0.34176)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 9 | 3
  CFB at Acute Follow-up: 145-168 hours | 0.2800 (0.39418) | -0.4533 (0.36295)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 9 | 3
  CFB at Extended Follow-up: Day 8 | 0.1900 (0.24850) | -0.2400 (0.72194)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 9 | 2
  CFB at Extended Follow-up: Day 15 | 0.1767 (0.41602) | -0.1100 (1.99404)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 7 | 1
  CFB at Extended Follow-up: Day 22 | 0.3029 (0.63746) | 1.7000
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 7 | 2
  CFB at Extended Follow-up: Day 29 | 0.0414 (0.21396) | 0.4850 (0.44548)

39. Primary Outcome: Change From Baseline in Hematology Parameter: Monocytes to Leukocytes Ratio Reported in Percentage of Cells
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, erythrocytes mean corpuscular hemoglobin concentration, erythrocytes mean corpuscular hemoglobin, erythrocytes mean corpuscular volume, erythrocytes, hematocrit, hemoglobin, leukocytes, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets. CFB in monocytes to leukocytes ratio is reported in terms of percentage of cells in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
percentage of cells
  Baseline: number analyzed (Participants) | 3 | 2
  Baseline | 7.67 (5.508) | 5.00 (4.243)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 2 | 1
  CFB at Infusion: 0-24 hours | 2.00 (0.000) | 1.00
  CFB at Infusion: 25-48 hours: number analyzed (Participants) | 2 | 1
  CFB at Infusion: 25-48 hours | -5.50 (7.778) | 13.00
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 3 | 1
  CFB at Infusion: 49-72 hours | -2.33 (0.577) | 15.00
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 2 | 1
  CFB at Infusion: 73-96 hours | -4.50 (4.950) | 8.00
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 2 | 1
  CFB at Infusion: 97-120 hours | -6.50 (9.192) | 8.00
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 2 | 1
  CFB at Acute Follow-up: 121-144 hours | -6.50 (9.192) | -1.00
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 2 | 1
  CFB at Acute Follow-up: 145-168 hours | -7.00 (9.899) | -2.00
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 2 | 0
  CFB at Extended Follow-up: Day 8 | -3.00 (8.485) |
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 2 | 0
  CFB at Extended Follow-up: Day 15 | -4.50 (6.364) |
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 2 | 1
  CFB at Extended Follow-up: Day 22 | -2.50 (4.950) | 0.00
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 2 | 0
  CFB at Extended Follow-up: Day 29 | -5.50 (9.192) |

40. Primary Outcome: Change From Baseline in Hematology Parameter: Neutrophil Levels
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, erythrocytes mean corpuscular hemoglobin concentration, erythrocytes mean corpuscular hemoglobin, erythrocytes mean corpuscular volume, erythrocytes, hematocrit, hemoglobin, leukocytes, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets. CFB in neutrophil levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
10^3 cells/uL
  Baseline: number analyzed (Participants) | 11 | 3
  Baseline | 7.957 (4.1505) | 13.863 (8.8017)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 10 | 3
  CFB at Infusion: 0-24 hours | 0.152 (2.4078) | -0.043 (1.7435)
  CFB at Infusion: 25-48 hours: number analyzed (Participants) | 10 | 3
  CFB at Infusion: 25-48 hours | -0.552 (3.1815) | -0.783 (2.9957)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 9 | 3
  CFB at Infusion: 49-72 hours | -1.406 (3.4517) | -0.167 (7.0002)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 9 | 3
  CFB at Infusion: 73-96 hours | -1.727 (3.6351) | -1.620 (6.0920)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 9 | 3
  CFB at Infusion: 97-120 hours | -0.743 (3.3970) | -2.653 (5.7315)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 9 | 3
  CFB at Acute Follow-up: 121-144 hours | -1.848 (4.2871) | -4.247 (6.7336)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 9 | 3
  CFB at Acute Follow-up: 145-168 hours | -1.440 (4.1338) | -3.517 (7.8465)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 9 | 3
  CFB at Extended Follow-up: Day 8 | -1.731 (4.4360) | -1.953 (7.7993)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 9 | 2
  CFB at Extended Follow-up: Day 15 | -2.372 (4.3518) | -9.825 (6.9650)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 7 | 2
  CFB at Extended Follow-up: Day 22 | -0.877 (3.2310) | -10.645 (7.9832)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 7 | 3
  CFB at Extended Follow-up: Day 29 | -1.590 (2.6196) | -6.323 (3.8800)

41. Primary Outcome: Change From Baseline in Hematology Parameter: Neutrophils to Leukocytes Ratio Reported in Percentage of Cells
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, erythrocytes mean corpuscular hemoglobin concentration, erythrocytes mean corpuscular hemoglobin, erythrocytes mean corpuscular volume, erythrocytes, hematocrit, hemoglobin, leukocytes, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets. CFB in neutrophils to leukocytes ratio is reported in terms of percentage of cells in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
percentage of cells
  Baseline: number analyzed (Participants) | 3 | 2
  Baseline | 75.67 (11.240) | 71.00 (8.485)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 2 | 1
  CFB at Infusion: 0-24 hours | -3.50 (9.192) | 19.00
  CFB at Infusion: 25-48 hours: number analyzed (Participants) | 2 | 1
  CFB at Infusion: 25-48 hours | 5.00 (5.657) | 6.00
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 3 | 1
  CFB at Infusion: 49-72 hours | 5.67 (10.504) | 3.00
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 2 | 1
  CFB at Infusion: 73-96 hours | 11.00 (11.314) | 2.00
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 2 | 1
  CFB at Infusion: 97-120 hours | 13.50 (17.678) | 9.00
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 2 | 1
  CFB at Acute Follow-up: 121-144 hours | 15.00 (14.142) | 31.00
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 2 | 1
  CFB at Acute Follow-up: 145-168 hours | 11.00 (8.485) | 25.00
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 2 | 0
  CFB at Extended Follow-up: Day 8 | 11.00 (11.314) |
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 2 | 0
  CFB at Extended Follow-up: Day 15 | 7.50 (9.192) |
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 2 | 1
  CFB at Extended Follow-up: Day 22 | -4.00 (7.071) | -10.00
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 2 | 0
  CFB at Extended Follow-up: Day 29 | 6.50 (14.849) |

42. Primary Outcome: Change From Baseline in Hematology Parameter: Platelet Levels
Description: Hematology measures included basophils, basophils to leukocytes ratio, eosinophils, eosinophils to leukocytes ratio, erythrocytes mean corpuscular hemoglobin concentration, erythrocytes mean corpuscular hemoglobin, erythrocytes mean corpuscular volume, erythrocytes, hematocrit, hemoglobin, leukocytes, lymphocytes, lymphocytes to leukocytes ratio, monocytes, monocytes to leukocytes ratio, neutrophils, neutrophils to leukocytes ratio, platelets. CFB in platelet levels is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
10^3 cells/uL
  Baseline: number analyzed (Participants) | 19 | 5
  Baseline | 260.76 (95.417) | 284.20 (80.707)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 18 | 5
  CFB at Infusion: 0-24 hours | 2.93 (68.821) | 21.40 (40.265)
  CFB at Infusion: 25-48 hours: number analyzed (Participants) | 19 | 5
  CFB at Infusion: 25-48 hours | 17.38 (92.854) | 34.40 (69.263)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 18 | 5
  CFB at Infusion: 49-72 hours | 21.59 (109.995) | 58.00 (95.533)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 18 | 5
  CFB at Infusion: 73-96 hours | 31.92 (112.963) | 77.80 (89.461)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 17 | 5
  CFB at Infusion: 97-120 hours | 57.49 (125.277) | 64.80 (101.043)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 17 | 5
  CFB at Acute Follow-up: 121-144 hours | 63.04 (138.415) | 61.80 (106.767)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 15 | 5
  CFB at Acute Follow-up: 145-168 hours | 81.98 (141.650) | 50.80 (130.555)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 15 | 4
  CFB at Extended Follow-up: Day 8 | 58.33 (120.436) | 48.75 (136.231)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 15 | 4
  CFB at Extended Follow-up: Day 15 | 153.89 (166.919) | 87.25 (177.265)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 13 | 4
  CFB at Extended Follow-up: Day 22 | 86.35 (204.827) | 49.75 (75.292)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 11 | 4
  CFB at Extended Follow-up: Day 29 | 25.76 (118.996) | 56.75 (112.512)

43. Primary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameter: Heart Rate
Description: ECG measures included heart rate, PR interval, QT interval, QRS duration and QTc interval. CFB in heart rate is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
beats/min
  Baseline: number analyzed (Participants) | 18 | 6
  Baseline | 84.3 (13.31) | 84.3 (19.64)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 16 | 6
  CFB at Infusion: 0-24 hours | -1.4 (16.87) | -6.8 (8.54)
  CFB at Infusion: 25-48 hours: number analyzed (Participants) | 16 | 6
  CFB at Infusion: 25-48 hours | -0.9 (16.58) | -1.2 (6.85)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 14 | 6
  CFB at Infusion: 49-72 hours | 10.9 (21.74) | -6.5 (22.28)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 15 | 6
  CFB at Infusion: 73-96 hours | 9.7 (15.49) | 7.7 (18.48)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 15 | 5
  CFB at Infusion: 97-120 hours | 15.9 (15.37) | 7.0 (19.62)
  CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 15 | 6
  CFB at Acute Follow-up: 121-144 hours | 13.2 (14.25) | 11.7 (22.76)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 14 | 6
  CFB at Acute Follow-up: 145-168 hours | 16.6 (16.91) | 17.0 (26.47)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 13 | 4
  CFB at Extended Follow-up: Day 8 | 19.2 (16.00) | 5.5 (22.87)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 12 | 4
  CFB at Extended Follow-up: Day 15 | 15.0 (23.09) | 5.5 (13.13)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 11 | 4
  CFB at Extended Follow-up: Day 22 | 13.8 (20.71) | 4.3 (26.73)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 9 | 4
  CFB at Extended Follow-up: Day 29 | 8.6 (13.60) | 7.0 (31.19)

44. Primary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters: PR Interval, QRS Interval, QT Interval and QTc Interval
Description: ECG measures included heart rate, PR interval, QT interval, QRS duration and QTc interval. CFB in PR interval, QT interval, QRS duration and QTc interval is reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: milliseconds (msec)
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
milliseconds (msec)
  PR interval: Baseline: number analyzed (Participants) | 18 | 6
  PR interval: Baseline | 151.0 [118 to 192] | 151.0 [132 to 182]
  PR interval: CFB at Infusion: 0-24 hours: number analyzed (Participants) | 16 | 6
  PR interval: CFB at Infusion: 0-24 hours | 2.0 [-40 to 10] | -2.0 [-16 to 18]
  PR interval: CFB at Infusion: 25-48 hours: number analyzed (Participants) | 16 | 6
  PR interval: CFB at Infusion: 25-48 hours | 3.0 [-40 to 148] | 3.0 [-4 to 15]
  PR interval: CFB at Infusion: 49-72 hours: number analyzed (Participants) | 14 | 5
  PR interval: CFB at Infusion: 49-72 hours | -13.0 [-42 to 16] | -2.0 [-8 to 18]
  PR interval: CFB at Infusion: 73-96 hours: number analyzed (Participants) | 15 | 5
  PR interval: CFB at Infusion: 73-96 hours | -2.0 [-22 to 22] | -4.0 [-6 to 7]
  PR interval: CFB at Infusion: 97-120 hours: number analyzed (Participants) | 15 | 5
  PR interval: CFB at Infusion: 97-120 hours | -12.0 [-32 to 68] | 2.0 [-22 to 26]
  PR interval: CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 15 | 6
  PR interval: CFB at Acute Follow-up: 121-144 hours | -8.0 [-25 to 23] | 3.5 [-28 to 12]
  PR interval: CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 14 | 6
  PR interval: CFB at Acute Follow-up: 145-168 hours | -11.0 [-38 to 14] | -2.0 [-26 to 24]
  PR interval: CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 13 | 3
  PR interval: CFB at Extended Follow-up: Day 8 | -10.0 [-30 to 4] | 0.0 [-20 to 2]
  PR interval: CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 12 | 4
  PR interval: CFB at Extended Follow-up: Day 15 | 0.0 [-54 to 26] | 4.0 [-16 to 18]
  PR interval: CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 11 | 4
  PR interval: CFB at Extended Follow-up: Day 22 | 2.0 [-26 to 36] | -6.5 [-40 to 10]
  PR interval: CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 9 | 4
  PR interval: CFB at Extended Follow-up: Day 29 | 2.0 [-20 to 14] | -8.0 [-18 to 22]
  QRS Interval: Baseline: number analyzed (Participants) | 18 | 6
  QRS Interval: Baseline | 85.0 [66 to 118] | 78.0 [40 to 100]
  QRS Interval: CFB at Infusion: 0-24 hours: number analyzed (Participants) | 16 | 6
  QRS Interval: CFB at Infusion: 0-24 hours | 1.0 [-12 to 14] | 1.5 [-4 to 20]
  QRS Interval: CFB at Infusion: 25-48 hours: number analyzed (Participants) | 16 | 6
  QRS Interval: CFB at Infusion: 25-48 hours | 0.0 [-14 to 40] | -1.0 [-8 to 6]
  QRS Interval: CFB at Infusion: 49-72 hours: number analyzed (Participants) | 14 | 6
  QRS Interval: CFB at Infusion: 49-72 hours | -3.0 [-20 to 6] | 2.0 [-2 to 5]
  QRS Interval: CFB at Infusion: 73-96 hours: number analyzed (Participants) | 15 | 6
  QRS Interval: CFB at Infusion: 73-96 hours | 0.0 [-16 to 18] | 0.0 [-6 to 20]
  QRS Interval: CFB at Infusion: 97-120 hours: number analyzed (Participants) | 15 | 5
  QRS Interval: CFB at Infusion: 97-120 hours | -4.0 [-32 to 14] | 0.0 [-14 to 20]
  QRS Interval: CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 15 | 6
  QRS Interval: CFB at Acute Follow-up: 121-144 hours | -2.0 [-32 to 8] | 0.0 [-14 to 20]
  QRS Interval: CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 14 | 6
  QRS Interval: CFB at Acute Follow-up: 145-168 hours | -6.0 [-28 to 16] | -3.0 [-94 to 20]
  QRS Interval: CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 13 | 4
  QRS Interval: CFB at Extended Follow-up: Day 8 | -2.0 [-28 to 0] | -3.5 [-16 to 0]
  QRS Interval: CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 12 | 4
  QRS Interval: CFB at Extended Follow-up: Day 15 | -5.0 [-47 to 6] | 2.0 [-2 to 40]
  QRS Interval: CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 11 | 4
  QRS Interval: CFB at Extended Follow-up: Day 22 | -4.0 [-26 to 6] | -1.0 [-4 to 20]
  QRS Interval: CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 9 | 4
  QRS Interval: CFB at Extended Follow-up: Day 29 | 2.0 [-26 to 12] | 5.0 [-4 to 40]
  QT Interval: Baseline: number analyzed (Participants) | 18 | 6
  QT Interval: Baseline | 363.0 [304 to 476] | 372.0 [280 to 462]
  QT Interval: CFB at Infusion: 0-24 hours: number analyzed (Participants) | 16 | 6
  QT Interval: CFB at Infusion: 0-24 hours | 19.5 [-84 to 200] | 24.5 [-26 to 49]
  QT Interval: CFB at Infusion: 25-48 hours: number analyzed (Participants) | 16 | 6
  QT Interval: CFB at Infusion: 25-48 hours | 19.5 [-102 to 236] | 3.0 [-40 to 30]
  QT Interval: CFB at Infusion: 49-72 hours: number analyzed (Participants) | 14 | 6
  QT Interval: CFB at Infusion: 49-72 hours | 1.0 [-168 to 238] | -14.0 [-66 to 144]
  QT Interval: CFB at Infusion: 73-96 hours: number analyzed (Participants) | 15 | 6
  QT Interval: CFB at Infusion: 73-96 hours | -4.0 [-62 to 128] | 0.0 [-76 to 118]
  QT Interval: CFB at Infusion: 97-120 hours: number analyzed (Participants) | 15 | 5
  QT Interval: CFB at Infusion: 97-120 hours | -34.0 [-164 to 72] | -36.0 [-102 to 66]
  QT Interval: CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 15 | 6
  QT Interval: CFB at Acute Follow-up: 121-144 hours | -28.0 [-168 to 238] | -32.0 [-126 to 40]
  QT Interval: CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 14 | 6
  QT Interval: CFB at Acute Follow-up: 145-168 hours | -32.0 [-164 to 74] | -34.0 [-156 to 18]
  QT Interval: CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 13 | 4
  QT Interval: CFB at Extended Follow-up: Day 8 | -36.0 [-186 to 42] | -35.0 [-138 to -6]
  QT Interval: CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 12 | 4
  QT Interval: CFB at Extended Follow-up: Day 15 | -32.0 [-176 to 72] | -8.0 [-116 to 16]
  QT Interval: CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 11 | 4
  QT Interval: CFB at Extended Follow-up: Day 22 | -28.0 [-132 to 51] | -22.0 [-102 to 24]
  QT Interval: CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 9 | 4
  QT Interval: CFB at Extended Follow-up: Day 29 | -28.0 [-132 to 29] | -63.0 [-96 to 80]
  QTc Interval: Baseline: number analyzed (Participants) | 18 | 6
  QTc Interval: Baseline | 435.5 [321 to 531] | 438.5 [393 to 454]
  QTc Interval: CFB at Infusion: 0-24 hours: number analyzed (Participants) | 16 | 6
  QTc Interval: CFB at Infusion: 0-24 hours | 7.5 [-55 to 219] | 7.0 [-58 to 42]
  QTc Interval: CFB at Infusion: 25-48 hours: number analyzed (Participants) | 16 | 6
  QTc Interval: CFB at Infusion: 25-48 hours | 11.5 [-49 to 277] | -12.5 [-59 to 29]
  QTc Interval: CFB at Infusion: 49-72 hours: number analyzed (Participants) | 14 | 6
  QTc Interval: CFB at Infusion: 49-72 hours | 3.5 [-103 to 275] | -14.0 [-38 to 36]
  QTc Interval: CFB at Infusion: 73-96 hours: number analyzed (Participants) | 15 | 6
  QTc Interval: CFB at Infusion: 73-96 hours | 8.0 [-30 to 145] | -13.5 [-41 to 152]
  QTc Interval: CFB at Infusion: 97-120 hours: number analyzed (Participants) | 15 | 5
  QTc Interval: CFB at Infusion: 97-120 hours | -2.0 [-88 to 106] | -17.0 [-38 to 43]
  QTc Interval: CFB at Acute Follow-up: 121-144 hours: number analyzed (Participants) | 15 | 6
  QTc Interval: CFB at Acute Follow-up: 121-144 hours | -12.0 [-87 to 319] | -9.0 [-31 to 10]
  QTc Interval: CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 14 | 6
  QTc Interval: CFB at Acute Follow-up: 145-168 hours | -4.0 [-96 to 93] | -17.5 [-52 to 15]
  QTc Interval: CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 13 | 4
  QTc Interval: CFB at Extended Follow-up: Day 8 | -15.0 [-111 to 83] | -54.5 [-86 to 14]
  QTc Interval: CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 11 | 4
  QTc Interval: CFB at Extended Follow-up: Day 15 | 2.0 [-104 to 71] | -6.5 [-50 to 3]
  QTc Interval: CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 10 | 4
  QTc Interval: CFB at Extended Follow-up: Day 22 | -8.5 [-57 to 51] | -33.5 [-37 to -14]
  QTc Interval: CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 8 | 4
  QTc Interval: CFB at Extended Follow-up: Day 29 | -2.0 [-72 to 51] | -19.0 [-51 to 23]

45. Primary Outcome: Number of Participants With Prior Anti-epileptic Drugs (AEDs) and Pressors Usage
Description: Prior AEDs and Pressors are those medications that ended before the initiation of SAGE-547 infusion.
Time Frame: Up to Day 29
Population: Safety population included all participants who were initiated with an infusion of SAGE-547.
Measure: Count of Participants; unit: Participants
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 19 | 6
Participants | 16 | 4

46. Secondary Outcome: Number of Participants With Relapse - Re-Initiation of Third-Line Agent
Description: Relapse of participants is defined as successfully weaning from a continuous IV third-line agent but subsequent requirement of re-initiation of a third-line agent following conclusion of SAGE-547 treatment.
Time Frame: Up to Day 29
Population: Efficacy population included all participants who completed the SAGE-547 infusion and who had at least one attempt to wean the third-line agent(s) before the start of the taper of the SAGE-547 infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 16 | 6
Participants | 5 | 1

47. Secondary Outcome: Number of Participants With Treatment Response (Treatment Responders)
Description: A responder was defined as a participant for whom it was not required to re-initiate continuous IV third-line therapy for refractory seizure control during the administration of SAGE-547 at the maintenance dose (prior to SAGE-547 taper infusion).
Time Frame: Up to 96 hours
Population: as for outcome 46
Measure: Count of Participants; unit: Participants
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 16 | 6
Participants | 13 | 4

48. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from the stop date/time of SAGE-547 maintenance to re-initiation of a third-line agent. If no re-initiation of a third-line agent was required, duration of response was not estimable and censored at Day 29 or death date, whichever occurred first. Kaplan-Meier method was used for the analysis.
Time Frame: Up to Day 29
Population: as for outcome 46
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 16 | 6
days | NA [NA to NA] — Median and confidence interval were not calculable due to more than 50% censored participants (8) in this treatment group. | NA [NA to NA] — Median and confidence interval were not calculable due to more than 50% censored participants (3) in this treatment group.

49. Secondary Outcome: Maximum Plasma Concentration (Cmax) of SAGE-547
Time Frame: Pre-dose (0 hours), 1, 2, 4, 8, 24, 48, 72, 96, 104, 112, 120 and 144 hours post-dose
Population: Pharmacokinetic (PK) population included all participants who received the study drug and had at least one PK sample taken. Overall number of participants analyzed is the number of participants with data available for analysis at the given time point for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 18 | 6
nanograms per milliliter (ng/mL) | 144.24 (65.263) | 200.82 (71.000)

50. Secondary Outcome: Time to Attain Maximum Observed Plasma Concentration (Tmax) of SAGE-547
Time Frame: Pre-dose (0 hours), 1, 2, 4, 8, 24, 48, 72, 96, 104, 112, 120 and 144 hours post-dose
Population: PK population included all participants who received the study drug and had at least one PK sample taken. Overall number of participants analyzed is the number of participants with data available for analysis at the given time point for this outcome measure.
Measure: Median (Full Range); unit: hours
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 18 | 6
hours | 1.010 [0.92 to 96.00] | 60.150 [0.93 to 118.52]

51. Secondary Outcome: Areas Under the Plasma SAGE-547 Concentration Time Curves From the Start of the Infusion Until the Time to the Last Sample (AUClast)
Time Frame: Pre-dose (0 hours), 1, 2, 4, 8, 24, 48, 72, 96, 104, 112, 120 and 144 hours post-dose
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: hour*nanograms per milliliter (h*ng/mL)
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 17 | 6
hour*nanograms per milliliter (h*ng/mL) | 7677.6 (2668.06) | 14260.0 (5048.01)

52. Secondary Outcome: Area Under the Plasma SAGE-547 Concentration-Time Curve in a 24 Hour Period (AUC24)
Time Frame: Pre-dose (0 hours), 1, 2, 4, 8 and 24 hours post-dose
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 18 | 6
h*ng/mL | 1590.3 (524.58) | 2728.3 (1010.14)

53. Secondary Outcome: Area Under the Plasma SAGE-547 Concentration-Time Curve (AUC1-96)
Time Frame: Pre-dose (0 hours), 1, 2, 4, 8, 24, 48, 72 and 96 hours post-dose
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 18 | 6
h*ng/mL | 6290.6 (2080.04) | 10801.7 (4006.70)

54. Secondary Outcome: Average Plasma Concentration (Cav) of SAGE-547
Time Frame: Pre-dose (0 hours), 1, 2, 4, 8, 24, 48, 72 and 96 hours post-dose
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 18 | 6
ng/mL | 66.22 (21.929) | 113.62 (42.079)

55. Secondary Outcome: Plasma Clearance (CL) of SAGE-547
Description: Clearance is defined as the volume of plasma from which a substance is completely removed per unit time.
Time Frame: Pre-dose (0 hours), 1, 2, 4, 8, 24, 48, 72, 96, 104, 112, 120 and 144 hours post-dose
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: liters per hour per kilogram (L/h/kg)
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 17 | 6
liters per hour per kilogram (L/h/kg) | 1.3999 (0.54525) | 1.2487 (0.65351)

56. Secondary Outcome: Change From Baseline in Modified Rankin Scale (mRS-9Q) Scores
Description: The mRS-9Q is a commonly used scale to determine disability and functional dependence due to neurological insult such as a stroke. It is a shortened version consisting of 9 questions. The score was categorized on the scale of 0 to 5 (0 = No symptoms, 1 = No significant disability, able to carry out all usual activities, despite some symptoms, 2 = Slight disability, able to look after own affairs without assistance, but unable to carry out all previous activities, 3 = Moderate disability, requires some help, but able to walk unassisted, 4 = Moderately severe disability, unable to attend to own bodily needs without assistance or unable to walk unassisted, and 5 = Severe disability, requires constant nursing care and attention, bedridden). Higher scores indicated worsening of symptoms.
Time Frame: Baseline (Screening) to Infusion at 49-72 hour, 73-96 hour; Extended follow-up at Day 8, 15, 22 and 29
Population: Efficacy population included all participants who completed the SAGE-547 infusion and who had at least one attempt to wean the third-line agent(s) before the start of the taper of the SAGE-547 infusion. Number analyzed is the number of participants with data available for analyses at the given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 16 | 6
score on a scale
  Baseline: number analyzed (Participants) | 16 | 5
  Baseline | 5.0 (0.00) | 5.0 (0.00)
  CBF at Infusion: 49-72 hours: number analyzed (Participants) | 16 | 5
  CBF at Infusion: 49-72 hours | 0.0 (0.00) | 0.0 (0.00)
  CFB at Infusion: 73-96 hours: number analyzed (Participants) | 16 | 5
  CFB at Infusion: 73-96 hours | 0.0 (0.00) | 0.0 (0.00)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 15 | 4
  CFB at Extended Follow-up: Day 8 | -0.1 (0.26) | 0.0 (0.00)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 15 | 4
  CFB at Extended Follow-up: Day 15 | -0.1 (0.35) | -0.3 (0.50)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 15 | 4
  CFB at Extended Follow-up: Day 22 | -0.4 (0.74) | -0.5 (0.58)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 13 | 4
  CFB at Extended Follow-up: Day 29 | -0.9 (1.50) | -1.0 (1.41)

57. Secondary Outcome: Change From Baseline in Clinical Global Impression: Severity Scale (CGI-S)
Description: The CGI-Severity (CGI-S) scale employs a 7-point Likert scale to assess the severity of participant's current illness state. Clinician responded to a question "Considering your total clinical experience with this particular population, how mentally ill is your patient at this time?" on the following scores: 1 = Normal, not at all ill, 2 = Borderline ill, 3 = Mildly ill, 4 = Moderately ill, 5 = Markedly ill, 6 = Severely ill, and 7 = Among the most extremely ill, where higher score = more affected.
Time Frame: Baseline (Screening), Extended follow-up at Days 8, 15, 22, and 29
Population: as for outcome 56
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 16 | 6
score on a scale
  Baseline | 6.9 (0.25) | 6.8 (0.41)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 15 | 5
  CFB at Extended Follow-up: Day 8 | -1.1 (1.06) | -1.2 (1.30)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 15 | 5
  CFB at Extended Follow-up: Day 15 | -2.3 (1.22) | -1.8 (1.79)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 15 | 5
  CFB at Extended Follow-up: Day 22 | -2.7 (1.63) | -2.4 (1.82)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 13 | 5
  CFB at Extended Follow-up: Day 29 | -3.0 (1.96) | -2.8 (2.39)

58. Secondary Outcome: Clinical Global Impression: Improvement Scale (CGI-I) Scores
Description: The CGI-I response was defined as having a score of 1 (very much improved) or 2 (much improved). CGI-I item employs a 7-point Likert scale to measure the overall improvement in the participant's condition post-treatment. The investigator rated the participant's total improvement whether or not it was due entirely to drug treatment. Response choices included: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse; where higher scores indicated worst outcomes. The CGI-I was only rated at post-treatment assessments. By definition, all CGI-I assessments were evaluated against baseline conditions.
Time Frame: Infusion at 0-24, 25-48, 49-72, 73-96, 97-120 hours; Acute follow-up at 121-144, 145-168 hours; Extended follow-up at Days 8, 15, 22 and 29
Population: as for outcome 56
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 16 | 6
score on a scale
  Infusion: 0-24 hours: number analyzed (Participants) | 16 | 5
  Infusion: 0-24 hours | 4.0 (0.37) | 4.0 (0.00)
  Infusion: 25-48 hours | 4.0 (0.52) | 4.5 (0.84)
  Infusion: 49-72 hours: number analyzed (Participants) | 16 | 5
  Infusion: 49-72 hours | 3.6 (0.81) | 3.6 (0.89)
  Infusion: 73-96 hours | 3.1 (0.81) | 3.7 (1.37)
  Infusion: 97-120 hours | 2.9 (0.81) | 3.0 (1.10)
  Acute Follow-up: 121-144 hours | 3.3 (1.30) | 4.0 (1.41)
  Acute Follow-up: 145-168 hours: number analyzed (Participants) | 16 | 5
  Acute Follow-up: 145-168 hours | 3.2 (1.52) | 3.2 (1.92)
  Extended Follow-up: Day 8: number analyzed (Participants) | 15 | 5
  Extended Follow-up: Day 8 | 2.9 (1.53) | 2.8 (1.10)
  Extended Follow-up: Day 15: number analyzed (Participants) | 15 | 5
  Extended Follow-up: Day 15 | 2.2 (1.21) | 2.4 (1.14)
  Extended Follow-up: Day 22: number analyzed (Participants) | 15 | 5
  Extended Follow-up: Day 22 | 2.3 (1.58) | 2.6 (1.95)
  Extended Follow-up: Day 29: number analyzed (Participants) | 13 | 5
  Extended Follow-up: Day 29 | 2.6 (1.89) | 2.4 (2.61)

59. Secondary Outcome: Change From Baseline in Glasgow Coma Scale (GCS) Scores
Description: The Glasgow Coma Scale is divided into three components which are scored separately: ocular response (assessment 1-4 points), motor response (assessment 1-6 points), verbal response (evaluation of 1-5 points). Scores for each component are added together to get the total score that will range between a minimum of 3 points (which corresponds to a participant who does not open his/her eyes and no motor response to stimulation or verbal response) and a maximum value of 15 points (corresponding to a participant with open eyes, obeying orders and maintaining a consistent language). It has been considered that the GCS score between 15 and 13 points corresponds to a slight alteration of consciousness, a score of 12-9 points with moderate impairment and 8 points or less with a serious deterioration in level of consciousness.
Time Frame: as for outcome 2
Population: as for outcome 56
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- SAGE-547 Standard Dose: Participants received SAGE-547 IV loading infusion of 286.6 μg/kg/hr for 1 hour on Day 1 followed by maintenance infusion of 86 μg/kg/hr for 95 hours from Days 1 to 4 followed by taper infusions of 64.5 μg/kg/hr, 43.0 μg/kg/hr, 21.5 μg/kg/hr at a duration of 8 hours each, on Day 5.
- SAGE-547 High Dose: Participants received SAGE-547 IV loading infusion of 286.6 μg/kg/hr for 1 hour on Day 1 followed by maintenance infusion A of 86 μg/kg/hr for 23 hours on Day 1 followed by maintenance infusion B of 156 μg/kg/hr for 72 hours from Days 2 to 4 followed by taper infusions of 125 μg/kg/hr, 94 μg/kg/hr, 62 μg/kg/hr, 31 μg/kg/hr at a duration of 6 hours each, on Day 5.
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 16 | 6
score on a scale
  Baseline | 3.9 (1.88) | 3.5 (1.22)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 16 | 5
  CFB at Infusion: 0-24 hours | -0.4 (1.26) | -0.2 (0.45)
  CFB at Infusion: 25-48 hours | -0.6 (1.63) | -0.5 (1.22)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 16 | 5
  CFB at Infusion: 49-72 hours | 0.9 (2.21) | 1.4 (1.34)
  CFB at Infusion: 73-96 hours | 1.1 (2.16) | 1.3 (2.42)
  CFB at Infusion: 97-120 hours | 2.4 (3.16) | 3.0 (3.69)
  CFB at Acute Follow-up: 121-144 hours | 3.3 (3.30) | 3.3 (3.93)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 16 | 5
  CFB at Acute Follow-up: 145-168 hours | 3.9 (3.98) | 5.0 (4.90)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 15 | 5
  CFB at Extended Follow-up: Day 8 | 3.9 (4.53) | 5.0 (4.90)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 15 | 5
  CFB at Extended Follow-up: Day 15 | 6.7 (4.73) | 5.4 (5.27)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 14 | 5
  CFB at Extended Follow-up: Day 22 | 6.9 (4.99) | 6.4 (4.83)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 12 | 5
  CFB at Extended Follow-up: Day 29 | 6.1 (5.70) | 7.4 (4.67)

60. Secondary Outcome: Change From Baseline in Richmond Agitation Sedation Scale (RASS) Score
Description: The RASS was an assessment of agitation and sedation in hospitalized participants, using a 10 point scale (ranged from -5 to +4), where, -5 = Unarousable, -4 = Deep sedation, -3 = Moderate sedation, -2 = Light sedation, -1 = Drowsy, 0 = Alert and calm, +1 = Restless, +2 = Agitated, +3 = Very agitated and +4 = Combative. Lower scores signify higher levels of sedation and higher scores signify heightened agitation. Participant in a calm and alert state would score a 0.
Time Frame: as for outcome 2
Population: as for outcome 56
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 16 | 6
score on a scale
  Baseline | -4.8 (0.54) | -4.8 (0.41)
  CFB at Infusion: 0-24 hours: number analyzed (Participants) | 16 | 5
  CFB at Infusion: 0-24 hours | -0.1 (0.25) | 0.0 (0.00)
  CFB at Infusion: 25-48 hours | -0.1 (0.44) | 0.0 (0.00)
  CFB at Infusion: 49-72 hours: number analyzed (Participants) | 16 | 5
  CFB at Infusion: 49-72 hours | 0.5 (1.32) | 0.8 (1.30)
  CFB at Infusion: 73-96 hours | 0.9 (1.41) | 0.7 (1.21)
  CFB at Infusion: 97-120 hours: number analyzed (Participants) | 15 | 6
  CFB at Infusion: 97-120 hours | 1.4 (1.59) | 1.3 (1.75)
  CFB at Acute Follow-up: 121-144 hours | 2.0 (1.97) | 1.3 (1.97)
  CFB at Acute Follow-up: 145-168 hours: number analyzed (Participants) | 16 | 5
  CFB at Acute Follow-up: 145-168 hours | 2.3 (2.24) | 1.4 (1.67)
  CFB at Extended Follow-up: Day 8: number analyzed (Participants) | 15 | 5
  CFB at Extended Follow-up: Day 8 | 2.3 (2.16) | 2.4 (2.61)
  CFB at Extended Follow-up: Day 15: number analyzed (Participants) | 15 | 5
  CFB at Extended Follow-up: Day 15 | 3.3 (1.79) | 2.2 (1.92)
  CFB at Extended Follow-up: Day 22: number analyzed (Participants) | 14 | 5
  CFB at Extended Follow-up: Day 22 | 3.4 (1.91) | 2.8 (2.17)
  CFB at Extended Follow-up: Day 29: number analyzed (Participants) | 12 | 5
  CFB at Extended Follow-up: Day 29 | 3.0 (2.22) | 2.8 (2.17)

61. Secondary Outcome: Number of Participants Who Survived
Description: Survival time was defined as duration of survival from screening up to Day 29.
Time Frame: Up to Day 29
Population: as for outcome 46
Measure: Count of Participants; unit: Participants
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
Number analyzed (Participants) | 16 | 6
Participants | 13 | 5

ADVERSE EVENTS:
Time Frame: Up to 29 days
Description: Safety Population included all participants who were initiated with an infusion of SAGE-547.
Arm/Group | SAGE-547 Standard Dose | SAGE-547 High Dose
All-Cause Mortality (participants affected / at risk) | 5/19 | 1/6
Serious Adverse Events (participants affected / at risk) | 14/19 | 2/6
Other Adverse Events (participants affected / at risk) | 15/19 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SAGE-547 Standard Dose (N=19) | SAGE-547 High Dose (N=6)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sepsis (Infections and infestations) | 1 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Tracheostomy infection (Infections and infestations) | 1 | 0
Chemical poisoning (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Convulsion (Nervous system disorders) | 2 | 0
Critical illness polyneuropathy (Nervous system disorders) | 1 | 0
Haemodynamic instability (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Obstructive shock (Vascular disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SAGE-547 Standard Dose (N=19) | SAGE-547 High Dose (N=6)
Urinary tract infection (Infections and infestations) | 1 | 2
Fungal skin infection (Infections and infestations) | 1 | 1
Oral candidiasis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 1 | 1
Pneumonia bacterial (Infections and infestations) | 2 | 0
Enterococcal infection (Infections and infestations) | 0 | 1
Paraspinal abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Bacterial tracheitis (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Candida infection (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Pneumonia pseudomonal (Infections and infestations) | 1 | 0
Urinary tract infection fungal (Infections and infestations) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Abdominal compartment syndrome (Gastrointestinal disorders) | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Lip dry (Gastrointestinal disorders) | 0 | 1
Swollen tongue (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Blood urea increased (Investigations) | 3 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 2
Lipase increased (Investigations) | 0 | 2
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood bicarbonate decreased (Investigations) | 0 | 1
ECG signs of myocardial ischaemia (Investigations) | 0 | 1
Glucose urine present (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Ammonia increased (Investigations) | 1 | 0
Blood albumin decreased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood chloride increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood phosphorus decreased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Carbon dioxide increased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Glomerular filtration rate decreased (Investigations) | 1 | 0
Haematocrit decreased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Monocyte count decreased (Investigations) | 1 | 0
Red blood cells urine positive (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 1 | 0
Hypotension (Vascular disorders) | 0 | 3
Hypertension (Vascular disorders) | 1 | 2
Deep vein thrombosis (Vascular disorders) | 2 | 1
Thrombosis (Vascular disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Oedema peripheral (General disorders) | 3 | 1
Pyrexia (General disorders) | 3 | 1
Hypothermia (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 2
Miliaria (Skin and subcutaneous tissue disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 2 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Haematuria (Renal and urinary disorders) | 3 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Nodal rhythm (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1
Pupils unequal (Eye disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can either be a party and subject to the same restrictions as the institution, or if not a party, the restrictions are described on the face of the contract (i.e., PI is a contractor of the institution; PI is part of a larger group of study personnel; institution has contracted with or otherwise bound all study personnel under confidentiality obligations and requirements to vest intellectual property to the institution).